CLINICAL TRIAL: NCT00144339
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group Trial Assessing the Rate of Decline of Lung Function With Tiotropium 18 mcg Inhalation Capsule Once Daily in Patients With Chronic Obstructive Pulmonary Disease (COPD).
Brief Title: Evaluation of the Long- Term Effects of Spiriva on Lung Function in COPD Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Model: Parallel | Purpose: Treatment
Other Study IDs: 205.235
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Results first posted 2009-08-17 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-04

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide

INTERVENTIONS:
Drug: tiotropium
Drug: placebo

SUMMARY:
The primary objective of this trial is to determine whether daily treatment with tiotropium (Spiriva®, Bromuro de Tiotropio®) inhalation capsule via HandiHaler® reduces the rate of decline in lung function over time in patients with COPD.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Male or female patients 40 years of age or older.
* Smoking history of at least 10 pack years.
* Diagnosis of COPD with post bronchodilator FEV1 less than or equal to 70% of predicted normal and FEV1<70% of FVC and on stable respiratory medication.

Exclusion Criteria:

* Significant diseases other than COPD which in the opinion of the investigator may put the patient at risk or influence the patients ability to participate.
* Myocardial infarction in past 6 months.
* Unstable or life threatening arrhythmia in past year.
* Hospitalization for NYHA heart failure class III or IV in past year.
* Active tuberculosis.
* Asthma.
* Pulmonary resection.
* Malignancy treated with radiation or chemotherapy in past 5 years.
* Respiratory infection in 4 weeks prior to screening.
* Known hypersensitivity to anticholinergic drugs or components.
* Known moderate to severe renal impairment.
* Known narrow angle glaucoma.
* Significant symptomatic BPH or bladder neck obstruction.
* Need for oxygen therapy >12 hr/day.
* Use of oral corticosteroids at unstable doses or >10 mg/day.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5993 (Actual)
Dates: Start 2002-12; Primary Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (490):
- United States (95):
  - 205.235.3779 Boehringer Ingelheim Investigational Site, Anniston, Alabama
  - 205.235.3785 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 205.235.3804 Boehringer Ingelheim Investigational Site, Jasper, Alabama
  - 205.235.3795 Boehringer Ingelheim Investigational Site, Mobile, Alabama
  - 205.235.3759 Boehringer Ingelheim Investigational Site, Phoenix, Arizona
  - 205.235.3770 Boehringer Ingelheim Investigational Site, Carmichael, California
  - 205.235.3778 Boehringer Ingelheim Investigational Site, Escondito, California
  - 205.235.3810 Boehringer Ingelheim Investigational Site, Lakewood, California
  - 205.235.3758 Boehringer Ingelheim Investigational Site, Long Beach, California
  - 205.235.3812 Boehringer Ingelheim Investigational Site, Long Beach, California
  - 205.235.3773 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 205.235.3800 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 205.235.3802 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 205.235.3786 Pulmonary and Critical Care Medicine, Orange, California
  - 205.235.3811 Boehringer Ingelheim Investigational Site, Palo Alto, California
  - 205.235.3741 Boehringer Ingelheim Investigational Site, Rancho Mirage, California
  - 205.235.3717 Boehringer Ingelheim Investigational Site, San Diego, California
  - 205.235.3781 Boehringer Ingelheim Investigational Site, San Diego, California
  - 205.235.3784 Boehringer Ingelheim Investigational Site, San Diego, California
  - 205.235.3760 Boehringer Ingelheim Investigational Site, Sepulveda, California
  - 205.235.3711 Boehringer Ingelheim Investigational Site, Stockton, California
  - 205.235.3764 Boehringer Ingelheim Investigational Site, Denver, Colorado
  - 205.235.3783 Boehringer Ingelheim Investigational Site, Wheat Ridge, Colorado
  - 205.235.3727 Boehringer Ingelheim Investigational Site, Hartford, Connecticut
  - 205.235.3808 Boehringer Ingelheim Investigational Site, Hartford, Connecticut
  - 205.235.3793 Boehringer Ingelheim Investigational Site, Norwalk, Connecticut
  - 205.235.3815 Boehringer Ingelheim Investigational Site, West Haven, Connecticut
  - 205.235.3706 Boehringer Ingelheim Investigational Site, Bay Pines, Florida
  - 205.235.3762 Boehringer Ingelheim Investigational Site, Brandon, Florida
  - 205.235.3707 Boehringer Ingelheim Investigational Site, Largo, Florida
  - 205.235.3703 Boehringer Ingelheim Investigational Site, Melbourne, Florida
  - 205.235.3775 Boehringer Ingelheim Investigational Site, Panama City, Florida
  - 205.235.3743 Boehringer Ingelheim Investigational Site, Sarasota, Florida
  - 205.235.3756 Boehringer Ingelheim Investigational Site, Tampa, Florida
  - 205.235.3739 Boehringer Ingelheim Investigational Site, West Palm Beach, Florida
  - 205.235.3719 Boehringer Ingelheim Investigational Site, Atlanta, Georgia
  - 205.235.3790 Boehringer Ingelheim Investigational Site, Atlanta, Georgia
  - 205.235.3716 Boehringer Ingelheim Investigational Site, Augusta, Georgia
  - 205.235.3794 Boehringer Ingelheim Investigational Site, Stockbridge, Georgia
  - 205.235.3724 Boehringer Ingelheim Investigational Site, Coeur d'Alene, Idaho
  - 205.235.3713 Boehringer Ingelheim Investigational Site, Normal, Illinois
  - 205.235.3768 Boehringer Ingelheim Investigational Site, Indianapolis, Indiana
  - 205.235.3749 Boehringer Ingelheim Investigational Site, Dubuque, Iowa
  - 205.235.3757 Boehringer Ingelheim Investigational Site, Olathe, Kansas
  - 205.235.3729 Boehringer Ingelheim Investigational Site, Lexington, Kentucky
  - 205.235.3737 Boehringer Ingelheim Investigational Site, Metairie, Louisiana
  - 205.235.3788 Boehringer Ingelheim Investigational Site, Shreveport, Louisiana
  - 205.235.3750 Boehringer Ingelheim Investigational Site, Bidderford, Maine
  - 205.235.3806 Boehringer Ingelheim Investigational Site, Baltimore, Maryland
  - 205.235.3721 Boehringer Ingelheim Investigational Site, Boston, Massachusetts
  - 205.235.3726 354 Birnie Ave, Springfield, Massachusetts
  - 205.235.3813 Boehringer Ingelheim Investigational Site, Ann Arbor, Michigan
  - 205.235.3732 Boehringer Ingelheim Investigational Site, Detroit, Michigan
  - 205.235.3809 Boehringer Ingelheim Investigational Site, Livonia, Michigan
  - 205.235.3751 Boehringer Ingelheim Investigational Site, Minneapolis, Minnesota
  - 205.235.3754 Boehringer Ingelheim Investigational Site, Minneapolis, Minnesota
  - 205.235.3789 Boehringer Ingelheim Investigational Site, Rochester, Minnesota
  - 205.235.3734 Boehringer Ingelheim Investigational Site, Chesterfield, Missouri
  - 205.235.3814 Boehringer Ingelheim Investigational Site, Kansas City, Missouri
  - 205.235.3747 Boehringer Ingelheim Investigational Site, St Louis, Missouri
  - 205.235.3763 Boehringer Ingelheim Investigational Site, Lebanon, New Hampshire
  - 205.235.3797 Boehringer Ingelheim Investigational Site, Cherry Hill, New Jersey
  - 205.235.3799 Boehringer Ingelheim Investigational Site, Summit, New Jersey
  - 205.235.3796 Boehringer Ingelheim Investigational Site, Albany, New York
  - 205.235.3807 Boehringer Ingelheim Investigational Site, Bay Shore, New York
  - 205.235.3765 Boehringer Ingelheim Investigational Site, Larchmont, New York
  - 205.235.3748 Boehringer Ingelheim Investigational Site, Mineola, New York
  - 205.235.3818 Boehringer Ingelheim Investigational Site, New York, New York
  - 205.235.3722 Boehringer Ingelheim Investigational Site, Rochester, New York
  - 205.235.3816 Boehringer Ingelheim Investigational Site, The Bronx, New York
  - 205.235.3730 Boehringer Ingelheim Investigational Site, Burlington, North Carolina
  - 205.235.3731 Boehringer Ingelheim Investigational Site, Chapel Hill, North Carolina
  - 205.235.3736 Boehringer Ingelheim Investigational Site, Durham, North Carolina
  - 205.235.3745 Boehringer Ingelheim Investigational Site, Elizabath City, North Carolina
  - 205.235.3712 Boehringer Ingelheim Investigational Site, Winston-Salem, North Carolina
  - 205.235.3723 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 205.235.3701 Boehringer Ingelheim Investigational Site, Cleveland, Ohio
  - 205.235.3791 Boehringer Ingelheim Investigational Site, Tulsa, Oklahoma
  - 205.235.3820 Boehringer Ingelheim Investigational Site, Portland, Oregon
  - 205.235.3725 Boehringer Ingelheim Investigational Site, Hershey, Pennsylvania
  - 205.235.3817 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - 205.235.3715 Boehringer Ingelheim Investigational Site, Providence, Rhode Island
  - 205.235.3803 Boehringer Ingelheim Investigational Site, El Paso, Texas
  - 205.235.3742 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 205.235.3787 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 205.235.3704 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 205.235.3752 Boehringer Ingelheim Investigational Site, Salt Lake City, Utah
  - 205.235.3744 Boehringer Ingelheim Investigational Site, Danville, Virginia
  - 205.235.3782 Boehringer Ingelheim Investigational Site, Fredericksburg, Virginia
  - 205.235.3771 Boehringer Ingelheim Investigational Site, Lynchburg, Virginia
  - 205.235.3738 Boehringer Ingelheim Investigational Site, Richmond, Virginia
  - 205.235.3792 Boehringer Ingelheim Investigational Site, Richmond, Virginia
  - 205.235.3761 Boehringer Ingelheim Investigational Site, Salem, Virginia
  - 205.235.3718 Boehringer Ingelheim Investigational Site, Spokane, Washington
  - 205.235.3780 Boehringer Ingelheim Investigational Site, La Crosse, Wisconsin
- Argentina (11):
  - 205.235.101, Buenos Aires
  - 205.235.101 Boehringer Ingelheim Investigational Site, Capital Federal
  - 205.235.103 Hospital Alemán, Capital Federal
  - 205.235.104 Hospital de Clinicas José de San Martín, Capital Federal
  - 205.235.105 Hospital General de Agudos José María Ramos Mejía, Capital Federal
  - 205.235.107 Policlínica Bancaria, Capital Federal
  - 205.235.108 Hospital General de Agudos Dr. Enrique Tornú, Capital Federal
  - 205.235.109 Hospital Muñiz, Capital Federal
  - 205.235.110 Hospital Privado - Centro Médico de Córdoba S.A., Parque Velez Sarlfield
  - 205.235.102 Instituto Cardiovascular de Rosario, Rosario
  - 205.235.106 Hospital Cetrángolo, Vicente López
- Australia (8):
  - 205.235.0205 Boehringer Ingelheim Investigational Site, Bankstown, New South Wales
  - 205.235.0202 Boehringer Ingelheim Investigational Site, Concord, New South Wales
  - 205.235.0209 Boehringer Ingelheim Investigational Site, Westmead, New South Wales
  - 205.235.0204 Boehringer Ingelheim Investigational Site, Cairns, Queensland
  - 205.235.0203 Boehringer Ingelheim Investigational Site, Redcliffe, Queensland
  - 205.235.0207 Boehringer Ingelheim Investigational Site, Port Lincoln, South Australia
  - 205.235.0206 Boehringer Ingelheim Investigational Site, Box Hill, Victoria
  - 205.235.0201 Boehringer Ingelheim Investigational Site, Geelong, Victoria
- Austria (5):
  - 205.235.0303 Boehringer Ingelheim Investigational Site, Graz
  - 205.235.0305 Boehringer Ingelheim Investigational Site, Innsbruck
  - 205.235.0304 Boehringer Ingelheim Investigational Site, Leoben
  - 205.235.0301 Boehringer Ingelheim Investigational Site, Vienna
  - 205.235.0302 Boehringer Ingelheim Investigational Site, Vienna
- Belgium (27):
  - 205.235.0439 Boehringer Ingelheim Investigational Site, Anderlecht
  - 205.235.0429 Boehringer Ingelheim Investigational Site, Baudour
  - 205.235.0421 Boehringer Ingelheim Investigational Site, Bruges
  - 205.235.0424 Boehringer Ingelheim Investigational Site, Brussels
  - 205.235.0432 Boehringer Ingelheim Investigational Site, Brussels
  - 205.235.0434 Boehringer Ingelheim Investigational Site, Brussels
  - 205.235.0422 Boehringer Ingelheim Investigational Site, Dendermonde
  - 205.235.0405 Boehringer Ingelheim Investigational Site, Edegem
  - 205.235.0414 Boehringer Ingelheim Investigational Site, Ghent
  - 205.235.0418 U.Z. Gent, Ghent
  - 205.235.0417 Boehringer Ingelheim Investigational Site, Herentals
  - 205.235.0402 Boehringer Ingelheim Investigational Site, Ieper
  - 205.235.0409 Boehringer Ingelheim Investigational Site, Kortrijk
  - 205.235.0407 Boehringer Ingelheim Investigational Site, Leuven
  - 205.235.0440 Boehringer Ingelheim Investigational Site, Luxembourg
  - 205.235.0403 Boehringer Ingelheim Investigational Site, Menen
  - 205.235.0406 Boehringer Ingelheim Investigational Site, Merksem
  - 205.235.0404 Boehringer Ingelheim Investigational Site, Middelheim
  - 205.235.0438 Boehringer Ingelheim Investigational Site, Mons
  - 205.235.0437 Boehringer Ingelheim Investigational Site, Namur
  - 205.235.0420 Boehringer Ingelheim Investigational Site, Neerpelt
  - 205.235.0435 Boehringer Ingelheim Investigational Site, Nobressart (attert)
  - 205.235.0423 Boehringer Ingelheim Investigational Site, Ostend
  - 205.235.0433 Boehringer Ingelheim Investigational Site, Tournai
  - 205.235.0412 Boehringer Ingelheim Investigational Site, Turnhout
  - 205.235.0413 Boehringer Ingelheim Investigational Site, Turnhout
  - 205.235.0428 Boehringer Ingelheim Investigational Site, Yvoir
- Brazil (14):
  - 205.235.510 Servico de Pneumologia, Florianópolis - SC
  - 205.235.508, Juiz de Fora - MG
  - 205.235.501, Porto Alegre - RS
  - 205.235.503, Porto Alegre - RS
  - 205.235.506, Porto Alegre - RS
  - 205.235.507 Depto.de Medicina Interna-Servico de pneumologia, Porto Alegre - RS
  - 205.235.502, Rio de Janeiro - RJ
  - 205.235.505 Dep.Medicina Especializada (DEMESP), Rio de Janeiro - RJ
  - 205.235.511 Departamento de Pneumologia, Salvador - BA
  - 205.235.504 ANEXO 2-Laboratório de Funcao Pulmonar, Santo André - SP
  - 205.235.512, São Paulo - SP
  - 205.235.513, São Paulo - SP
  - 205.235.514 Unidade de Coracao e Pulmao do Dto. de Medicina, São Paulo - SP
  - 205.235.515 Lar Escola São Francisco / Setor de Pneumologia, São Paulo - SP
- Czechia (26):
  - 205.235.0712 Boehringer Ingelheim Investigational Site, Benešov
  - 205.235.0711 Boehringer Ingelheim Investigational Site, Beroun
  - 205.235.0718 Clinic of Functional Diagnostics and Rehabilitation, Brno
  - 205.235.0725 University Hospital Brno, Brno
  - 205.235.0720 Office of Pulmonology and Respiratory Diseases, Český Těšín
  - 205.235.0717 Pulmonary Clinic, Hradec Králové
  - 205.235.0705 Boehringer Ingelheim Investigational Site, Jablonec nad Nisou
  - 205.235.0726 Private Office of Pulmonary Diseases, Jaroměř
  - 205.235.0722 Hospital Kromeriz, Kroměříž
  - 205.235.0724 District Hospital Kyjov, Kyjov
  - 205.235.0704 Boehringer Ingelheim Investigational Site, Lovosice
  - 205.235.0702 Boehringer Ingelheim Investigational Site, Mariánské Lázně
  - 205.235.0701 Boehringer Ingelheim Investigational Site, Pilsen
  - 205.235.0703 Boehringer Ingelheim Investigational Site, Pilsen
  - 205.235.0706 Boehringer Ingelheim Investigational Site, Prague
  - 205.235.0707 Boehringer Ingelheim Investigational Site, Prague
  - 205.235.0709 Boehringer Ingelheim Investigational Site, Prague
  - 205.235.0710 Boehringer Ingelheim Investigational Site, Prague
  - 205.235.0715 Boehringer Ingelheim Investigational Site, Prague
  - 205.235.0708 Boehringer Ingelheim Investigational Site, Praha 5 - Nove Butovice
  - 205.235.0723 Office of Pulmonary and Respiratory Diseases, Přerov
  - 205.235.0721 Office of Pulmonary Diseases, Příbor
  - 205.235.0713 Boehringer Ingelheim Investigational Site, Strakonice
  - 205.235.0714 Boehringer Ingelheim Investigational Site, Tábor
  - 205.235.0719 Office of Pulmonology and Respiratory Diseases, Ústí nad Orlicí
  - 205.235.0716 Boehringer Ingelheim Investigational Site, Znojmo
- Denmark (29):
  - 205.235.0804 Boehringer Ingelheim Investigational Site, Aalborg
  - 205.235.0826 Boehringer Ingelheim Investigational Site, Aalborg SV
  - 205.235.0803 Boehringer Ingelheim Investigational Site, Aarhus
  - 205.235.0831 Boehringer Ingelheim Investigational Site, Copenhagen
  - 205.235.0828 Boehringer Ingelheim Investigational Site, Copenhagen K
  - 205.235.0802 Boehringer Ingelheim Investigational Site, Copenhagen NV
  - 205.235.0816 Boehringer Ingelheim Investigational Site, Elsinore
  - 205.235.0807 Boehringer Ingelheim Investigational Site, Fåborg
  - 205.235.0821 Boehringer Ingelheim Investigational Site, Frederikshavn
  - 205.235.0832 Boehringer Ingelheim Investigational Site, Frederikssund
  - 205.235.0805 Boehringer Ingelheim Investigational Site, Hellerup
  - 205.235.0835 Boehringer Ingelheim Investigational Site, Hellerup
  - 205.235.0811 Boehringer Ingelheim Investigational Site, Hillerød
  - 205.235.0834 Boehringer Ingelheim Investigational Site, Hobro
  - 205.235.0806 Boehringer Ingelheim Investigational Site, Holbæk
  - 205.235.0814 Boehringer Ingelheim Investigational Site, Holstebro
  - 205.235.0801 Boehringer Ingelheim Investigational Site, Hvidovre
  - 205.235.0833 Boehringer Ingelheim Investigational Site, Kalundborg
  - 205.235.0830 Boehringer Ingelheim Investigational Site, Kolding
  - 205.235.0819 Boehringer Ingelheim Investigational Site, Nykøbing Falster
  - 205.235.0810 Boehringer Ingelheim Investigational Site, Næstved
  - 205.235.0809 Boehringer Ingelheim Investigational Site, Odense C
  - 205.235.0815 Boehringer Ingelheim Investigational Site, Randers
  - 205.235.0824 Boehringer Ingelheim Investigational Site, Silkeborg
  - 205.235.0813 Boehringer Ingelheim Investigational Site, Skive
  - 205.235.0822 Boehringer Ingelheim Investigational Site, Skive
  - 205.235.0820 Boehringer Ingelheim Investigational Site, Slagelse
  - 205.235.0808 Boehringer Ingelheim Investigational Site, Svendborg
  - 205.235.0827 Boehringer Ingelheim Investigational Site, Værløse
- Finland (5):
  - 205.235.0903 Boehringer Ingelheim Investigational Site, Helsinki
  - 205.235.0901 Boehringer Ingelheim Investigational Site, Jyväskylä
  - 205.235.0905 Boehringer Ingelheim Investigational Site, Kotka
  - 205.235.0904 Boehringer Ingelheim Investigational Site, Lahti
  - 205.235.0902 Boehringer Ingelheim Investigational Site, Pori
- France (17):
  - 205.235.1004 Clinique Toulouse Lautrec, Albi
  - 205.235.1007 Cabinet Médical, Albi
  - 205.235.1015 Centre Hospitalier, Barbezieux-Saint-Hilaire
  - 205.235.1012 Cabinet Médical, Bourges
  - 205.235.1024 Cabinet Médical, Chamalières
  - 205.235.1006 Centre Hospitalier de Chauny, Chauny
  - 205.235.1005 Polyclinique, Cholet
  - 205.235.1013 Cabinet Médical, La Teste-de-Buch
  - 205.235.1020 Cabinet Médical, Marseille
  - 205.235.1023 Cabinet Médical, Montauban
  - 205.235.1025 Centre Médical Erdre Saint Augustin, Nantes
  - 205.235.1002 Cabinet médical, Nice
  - 205.235.1001 Hôpital Bichat, Paris
  - 205.235.1016 Cabinet Médical, Provins
  - 205.235.1019 Cabinet Médical, Strasbourg
  - 205.235.1009 Centre Hospitalier de Bigorre, Tarbes
  - 205.235.1021 Clinique Pasteur, Toulouse
- Germany (14):
  - 205.235.1113 Boehringer Ingelheim Investigational Site, Berlin
  - 205.235.1114 Boehringer Ingelheim Investigational Site, Berlin
  - 205.235.1103 Boehringer Ingelheim Investigational Site, Brake
  - 205.235.1105 Boehringer Ingelheim Investigational Site, Braunschweig
  - 205.235.1104 Boehringer Ingelheim Investigational Site, Bruchsal
  - 205.235.1115 Boehringer Ingelheim Investigational Site, Hanover
  - 205.235.1109 Boehringer Ingelheim Investigational Site, Kaufbeuren
  - 205.235.1108 Boehringer Ingelheim Investigational Site, Loerrach
  - 205.235.1102 Boehringer Ingelheim Investigational Site, Lübeck
  - 205.235.1106 Boehringer Ingelheim Investigational Site, München
  - 205.235.1110 Boehringer Ingelheim Investigational Site, München
  - 205.235.1101 Boehringer Ingelheim Investigational Site, Ulm
  - 205.235.1107 Boehringer Ingelheim Investigational Site, Weyhe
  - 205.235.1112 Boehringer Ingelheim Investigational Site, Wiesloch
- Greece (10):
  - 205.235.1202 8th Pulmonology Clinic "Sotiria" Athens Chest Hospital, Athens
  - 205.235.1203 Boehringer Ingelheim Investigational Site, Athens
  - 205.235.1201 Boehringer Ingelheim Investigational Site, Heraklion
  - 205.235.1211 Boehringer Ingelheim Investigational Site, Kavala
  - 205.235.1204 Boehringer Ingelheim Investigational Site, Larissa
  - 205.235.1209 Boehringer Ingelheim Investigational Site, Pátrai
  - 205.235.1210 Boehringer Ingelheim Investigational Site, Pátrai
  - 205.235.1205 Boehringer Ingelheim Investigational Site, Thessaloniki
  - 205.235.1206 Boehringer Ingelheim Investigational Site, Thessaloniki
  - 205.235.1207 Boehringer Ingelheim Investigational Site, Thessaloniki
- Hong Kong (4):
  - 205.235.1401 Boehringer Ingelheim Investigational Site, Hong Kong
  - 205.235.1403 Boehringer Ingelheim Investigational Site, Hong Kong
  - 205.235.1402 Boehringer Ingelheim Investigational Site, Kowloon
  - 205.235.1404 Boehringer Ingelheim Investigational Site, Kowloon
- Hungary (20):
  - 205.235.1303 Boehringer Ingelheim Investigational Site, Budapest
  - 205.235.1308 Boehringer Ingelheim Investigational Site, Budapest
  - 205.235.1309 Boehringer Ingelheim Investigational Site, Budapest
  - 205.235.1310 Boehringer Ingelheim Investigational Site, Budapest
  - 205.235.1311 Boehringer Ingelheim Investigational Site, Budapest
  - 205.235.1318 Boehringer Ingelheim Investigational Site, Debrecen
  - 205.235.1314 Boehringer Ingelheim Investigational Site, Deszk
  - 205.235.1306 Boehringer Ingelheim Investigational Site, Érd
  - 205.235.1315 Boehringer Ingelheim Investigational Site, Farkasgyepü
  - 205.235.1320 Boehringer Ingelheim Investigational Site, Gyula
  - 205.235.1307 Boehringer Ingelheim Investigational Site, Kiskunhalas
  - 205.235.1304 Boehringer Ingelheim Investigational Site, Miskolc
  - 205.235.1317 Boehringer Ingelheim Investigational Site, Mosonmagyaróvár
  - 205.235.1301 Boehringer Ingelheim Investigational Site, Pécs
  - 205.235.1313 Boehringer Ingelheim Investigational Site, Solymár
  - 205.235.1305 Boehringer Ingelheim Investigational Site, Sopron
  - 205.235.1319 Boehringer Ingelheim Investigational Site, Szombathely
  - 205.235.1302 Boehringer Ingelheim Investigational Site, Tatabánya
  - 205.235.1316 Boehringer Ingelheim Investigational Site, Törökbálint
  - 205.235.1312 Boehringer Ingelheim Investigational Site, Veszprém
- Ireland (3):
  - 205.235.1501 Boehringer Ingelheim Investigational Site, Dublin
  - 205.235.1503 Boehringer Ingelheim Investigational Site, Dublin
  - 205.235.1505 Boehringer Ingelheim Investigational Site, Dublin
- Italy (31):
  - 205.235.1631 A. O. SS. Antonio e Biagio e Arrigo, Alessandria
  - 205.235.1613 A. O. S. Giuseppe Moscati, Avellino
  - 205.235.1618 Ospedale Bellaria, Bologna
  - 205.235.1649 Ospedale di Circolo di Busto Arsizio, Busto Arsizio (VA)
  - 205.235.1635 P. O. Roberto Binaghi, Cagliari
  - 205.235.1623 A. O. di Carrara, Carrara (Massa)
  - 205.235.1645 Ospedale Civile "Zappatoni", Cassano D'adda (Milano)
  - 205.235.1617 Ospedale S. Camillo De Lellis, Chieti
  - 205.235.1612 A. O. S. Antonio Abate, Erice (Trapani)
  - 205.235.1622 A. O. S. Anna, Ferrara
  - 205.235.1646 A. O. di Careggi, Florence
  - 205.235.1647 A. O. Careggi, Florence
  - 205.235.1615 Ospedale S. Martino, Genova
  - 205.235.1603 P. O. di Gubbio, Gubbio (Perugia)
  - 205.235.1619 A. O. Fratelli Crobu, Iglesias (Cagliari)
  - 205.235.1648 Ospedale "S. Maria di Collemaggio", L’Aquila
  - 205.235.1624 Ospedale di Macerata, Macerata
  - 205.235.1634 P. O. Luigi Sacco, Milan
  - 205.235.1639 Ospedale Maggiore, Modica (Ragusa)
  - 205.235.1629 A. O. S. Luigi Gonzaga, Orbassano (Torino)
  - 205.235.1604 P. O. R. Silvestrini, Perugia
  - 205.235.1601 Presidio Ospedaliero di Cisanello, Pisa
  - 205.235.1643 A. O. Santa Maria degli Angeli, Pordenone
  - 205.235.1614 Ospedale Misericordia e Dolce, Prato
  - 205.235.1607 Università degli Studi di Sassari, Sassari
  - 205.235.1608 ASL 1 di Sassari, Sassari
  - 205.235.1606 ASL 4 di Terni, Terni
  - 205.235.1632 ASL 4 - Distretto 2, Torino
  - 205.235.1633 A. O. Umberto I, Torrette Di Ancona (Ancona)
  - 205.235.1640 P. O. Cà Foncello, Treviso
  - 205.235.1602 Ospedale di Voghera, Voghera (Pavia)
- Japan (12):
  - 205.235.1706 Juntendo University Hospital, Bunkyo-ku, Tokyo
  - 205.235.1705 Kameda Medical Center, Kamogawa, Chiba
  - 205.235.1713 Komaki City Hospital, Komaki, Aichi
  - 205.235.1712 Kurume University Hospital, Kurume, Fukuoka
  - 205.235.1708 Shinshu University, Matsumoto, Nagano
  - 205.235.1702 Iwate Medical University Hospital, Morioka, Iwate
  - 205.235.1710 Osaka City University Hospital, Osaka, Osaka
  - 205.235.1711 Kinki University Hospital, Osakasayama, Osaka
  - 205.235.1701 Hokkaido University, Sapporo, Hokkaido
  - 205.235.1703 Tohoku University Hospital, Sendai, Miyagi
  - 205.235.1709 Tosei General Hospital, Seto, Aichi
  - 205.235.1704 Hiraka General Hospital, Yokote, Akita
- Lithuania (3):
  - 205.235.1801 Boehringer Ingelheim Investigational Site, Kaunas
  - 205.235.1802 Boehringer Ingelheim Investigational Site, Kaunas
  - 205.235.1803 Boehringer Ingelheim Investigational Site, Vilnius
- Malaysia (3):
  - 205.235.1901 Boehringer Ingelheim Investigational Site, Kuala Lumpur
  - 205.235.1902 Boehringer Ingelheim Investigational Site, Kuala Lumpur
  - 205.235.1903 Boehringer Ingelheim Investigational Site, Kuala Lumpur
- Mexico (7):
  - 205.235.2004 Edif. Dr. Rodrigo F. Barragan, P.B., Col. Mitras Centro, Monterrey, N.L.
  - 205.235.2002, Guadalajara, Jal.
  - 205.235.2005, Mexico City
  - 205.235.2006 Tlalpan 4000, Pabellón 5, EPOC, Mexico City
  - 205.235.2009, Puebla City
  - 205.235.2010 Depto. De Ivestigación, Toluca
  - 205.235.2003, Zapopan, Jalisco
- Netherlands (13):
  - 205.235.2110 Poli Longziekten, Almelo
  - 205.235.2105 Lokatie De Lichtenberg, Amersfoort
  - 205.235.2107 Poli Longziekten, Delft
  - 205.235.2106 Lokatie Dordwijk, Dordrecht
  - 205.235.2104 Poli longziekten, Eindhoven
  - 205.235.2102 Martini Ziekenhuis Groningen, Groningen
  - 205.235.2112 Poli Longziekten, Harderwijk
  - 205.235.2115 Poli Longziekten, Heerenveen
  - 205.235.2101 Atrium medisch centrum, Heerlen
  - 205.235.2114 Poli Longziekten, Hengelo
  - 205.235.2108 Poli Longziekten, Leeuwarden
  - 205.235.2109 Poli Longziekten, Rotterdam
  - 205.235.2111 Antonius Ziekenhuis, Sneek
- New Zealand (2):
  - 205.235.0211 Boehringer Ingelheim Investigational Site, Auckland
  - 205.235.0212 Boehringer Ingelheim Investigational Site, Christchurch, New Zealand
- Norway (4):
  - 205.235.2202 Boehringer Ingelheim Investigational Site, Arendal
  - 205.235.2201 Boehringer Ingelheim Investigational Site, Fredrikstad
  - 205.235.2205 Boehringer Ingelheim Investigational Site, Sandvika
  - 205.235.2204 Boehringer Ingelheim Investigational Site, Straume
- Philippines (5):
  - 205.235.2301 Philippine General Hospital, Manila
  - 205.235.2305 University of Santo Tomas Hospital, Manila
  - 205.235.2302 Philippine Heart Center, Quezon City
  - 205.235.2303 Veterans Memorial Medical Center, Quezon City
  - 205.235.2304 Lung Center of the Philippines, Quezon City
- Poland (10):
  - 205.235.2410 Boehringer Ingelheim Investigational Site, Gdansk
  - 205.235.2407 Boehringer Ingelheim Investigational Site, Katowice
  - 205.235.2408 Boehringer Ingelheim Investigational Site, Krakow
  - 205.235.2405 Boehringer Ingelheim Investigational Site, Lodz
  - 205.235.2409 Boehringer Ingelheim Investigational Site, Lodz
  - 205.235.2401 Boehringer Ingelheim Investigational Site, Warsaw
  - 205.235.2402 Boehringer Ingelheim Investigational Site, Warsaw
  - 205.235.2403 Boehringer Ingelheim Investigational Site, Warsaw
  - 205.235.2404 Boehringer Ingelheim Investigational Site, Wroclaw
  - 205.235.2406 Boehringer Ingelheim Investigational Site, Zabrze
- Portugal (5):
  - 205.235.2504 Centro Hospitalar de Coimbra, Coimbra
  - 205.235.2503 Hospital Pulido Valente, Lisbon
  - 205.235.2505 Hospital de Santa Marta, Lisbon
  - 205.235.2501 Hospital de São João, Porto
  - 205.235.2502 Centro Hospitalar de Vila Nova de Gaia, Vila Nova de Gaia
- Russia (5):
  - 205.235.2601 Boehringer Ingelheim Investigational Site, Moscow
  - 205.235.2602 Boehringer Ingelheim Investigational Site, Moscow
  - 205.235.2603 Boehringer Ingelheim Investigational Site, Moscow
  - 205.235.2605 Boehringer Ingelheim Investigational Site, Moscow
  - 205.235.2604 Boehringer Ingelheim Investigational Site, Saint Petersburg
- Singapore (3):
  - 205.235.1904 Boehringer Ingelheim Investigational Site, Singapore
  - 205.235.1905 Boehringer Ingelheim Investigational Site, Singapore
  - 205.235.1906 Boehringer Ingelheim Investigational Site, Singapore
- Slovakia (5):
  - 205.235.2701 Boehringer Ingelheim Investigational Site, Bratislava
  - 205.235.2702 Boehringer Ingelheim Investigational Site, Bratislava
  - 205.235.2703 Boehringer Ingelheim Investigational Site, Martin
  - 205.235.2704 Boehringer Ingelheim Investigational Site, Poprad
  - 205.235.2705 Boehringer Ingelheim Investigational Site, Topoľčany
- Slovenia (5):
  - 205.235.2801 Boehringer Ingelheim Investigational Site, Golnik
  - 205.235.2802 Boehringer Ingelheim Investigational Site, Golnik
  - 205.235.2805 Boehringer Ingelheim Investigational Site, Kamnik
  - 205.235.2803 Boehringer Ingelheim Investigational Site, Ljubljana
  - 205.235.2804 Boehringer Ingelheim Investigational Site, Topolšica
- South Africa (11):
  - 205.235.2908, Bloemfontein
  - 205.235.2910, Cape Town
  - 205.235.2912, Cape Town
  - 205.235.2904, Durban
  - 205.235.2911, Durban
  - 205.235.2902, George
  - 205.235.2905, Paarl
  - 205.235.2901 Boehringer Ingelheim Investigational Site, Pretoria
  - 205.235.2906, Somerset West
  - 205.235.2903, Vanderbijlpark
  - 205.235.2909, Welkom
- Spain (36):
  - 205.235.3014 Complejo Hospitalario Juan Canalejo, A Coruña
  - 205.235.3026 Hospital General Universitario de Alicante, Alicante
  - 205.235.3011 Complejo Hospitalario Infanta Cristina, Badajoz
  - 205.235.3006 Hospital Germans Trias i Pujol, Badalona (Barcelona)
  - 205.235.3022 Hospital de Cruces, Barakaldo (Bilbao)
  - 205.235.3003 Hospital Clínic i Provincial de Barcelona, Barcelona
  - 205.235.3008 Hospital Vall d'Hebrón, Barcelona
  - 205.235.3023 Hospital Dr. Josep Trueta, Girona
  - 205.235.3004 Hospital General Universitario de Guadalajara, Guadalajara
  - 205.235.3005 Hospital General San Jorge de Huesca, Huesca
  - 205.235.3021 Hospital de Jerez de la Frontera, Jerez de la Frontera
  - 205.235.3010 Hospital Severo Ochoa, Leganés, Madrid
  - 205.235.3009 Hospital Clínico San Carlos, Madrid
  - 205.235.3013 Clínica Puerta de Hierro, Madrid
  - 205.235.3017 Hospital Ramón y Cajal, Madrid
  - 205.235.3020 Hospital Universitario La Paz, Madrid
  - 205.235.3028 Hospital Universitario de la Princesa, Madrid
  - 205.235.3031 Hospital Gregorio Marañón, Madrid
  - 205.235.3036 Hospital 12 de Octubre, Madrid
  - 205.235.3033 Hospital General Carlos Haya, Málaga
  - 205.235.3027 Complejo Asistencial Son Dureta, Palma de Mallorca
  - 205.235.3024 Hospital de Montecelo, Pontevedra
  - 205.235.3016 Hospital Universitari de Sant Joan, Reus (Tarragona)
  - 205.235.3015 Corporació Sanitaria Parc Taulí de Sabadell, Sabadell (Barcelona)
  - 205.235.3037 Hsopital Universitario Ntra. Sra. de la Candelaria, Santa Cruz de Tenerife
  - 205.235.3039 Hospital Universitario Marqués de Valdecilla, Santander
  - 205.235.3019 Hospital Vírgen de la Macarena, Seville
  - 205.235.3035 Hospital Universitario Vírgen del Rocío, Seville
  - 205.235.3001 Hospital Mutua Terrassa, Terrassa (Barcelona)
  - 205.235.3002 Hospital Clínico Universitario de Valencia, Valencia
  - 205.235.3025 Hospital Universitario Dr. Peset, Valencia
  - 205.235.3032 Hospital Arnau de Vilanova, Valencia
  - 205.235.3034 Hospital La Fe, Valencia
  - 205.235.3018 Complejo Hospitalario Xeral - Cíes, Vigo
  - 205.235.3030 Hospital Miguel Servet, Zaragoza
  - 205.235.3038 Hospital Clínico Lozano Blesa, Zaragoza
- Switzerland (7):
  - 205.235.3202 Boehringer Ingelheim Investigational Site, Basel
  - 205.235.3203 Universitätsspital Basel, Basel
  - 205.235.3204 Boehringer Ingelheim Investigational Site, Faltigberg
  - 205.235.3205 Boehringer Ingelheim Investigational Site, Lugano
  - 205.235.3206 Boehringer Ingelheim Investigational Site, Montana
  - 205.235.3208 Boehringer Ingelheim Investigational Site, Winterthur
  - 205.235.3201 Boehringer Ingelheim Investigational Site, Zurich
- Taiwan (3):
  - 205.235.3301 Boehringer Ingelheim Investigational Site, Taipei
  - 205.235.3302 Boehringer Ingelheim Investigational Site, Taipei
  - 205.235.3303 Boehringer Ingelheim Investigational Site, Taipei
- Thailand (5):
  - 205.235.3402 Boehringer Ingelheim Investigational Site, Bangkok
  - 205.235.3403 Boehringer Ingelheim Investigational Site, Bangkok
  - 205.235.3404 Boehringer Ingelheim Investigational Site, Bangkok
  - 205.235.3401 Boehringer Ingelheim Investigational Site, Chiang Mai
  - 205.235.3405 Boehringer Ingelheim Investigational Site, Khon Kaen
- Turkey (Türkiye) (12):
  - 205.235.3510 Cukurova Tip Fakultesi Balcali Hastanesi, Adana
  - 205.235.3506 Hacettepe Tip Fakultesi, Ankara
  - 205.235.3507 Ankara SSK Diskapi Egitim Hastanesi, Ankara
  - 205.235.3508 Atatürk Gögüs Hastaliklari ve Gögüs Cerrahi, Ankara
  - 205.235.3509 Atatürk Üniversitesi Tip Fakultesi Aziziye, Erzurum
  - 205.235.3511 Osmangazi Universitesi Tip Fakültesi, Eskişehir
  - 205.235.3501 Istanbul Universitesi Cerrahpasa Tip Fakultesi, Istanbul
  - 205.235.3502 Yedikule Gögüs Hastaliklari Hastanesi, Istanbul
  - 205.235.3503 Tophanelioglu Cad. No: 13/15, Istanbul
  - 205.235.3504 Cevizli E5 Karayolu, Istanbul
  - 205.235.3505 Istanbul Universitesi Tip Fakültesi, Istanbul
  - 205.235.3512 DokuzEylül Universitesi Tip Fakultesi Gögüs Hastaliklari ABD, Izmir
- United Kingdom (15):
  - 205.235.3615 Boehringer Ingelheim Investigational Site, Aberdeen
  - 205.235.3611 Boehringer Ingelheim Investigational Site, Chertsey
  - 205.235.3613 Boehringer Ingelheim Investigational Site, Chesterfield
  - 205.235.3608 Boehringer Ingelheim Investigational Site, Cottingham, Hull
  - 205.235.3605 Boehringer Ingelheim Investigational Site, Exeter
  - 205.235.3602 Boehringer Ingelheim Investigational Site, Glasgow
  - 205.235.3610 Boehringer Ingelheim Investigational Site, Leeds
  - 205.235.3607 Boehringer Ingelheim Investigational Site, Leicester
  - 205.235.3604 Boehringer Ingelheim Investigational Site, Middleton
  - 205.235.3612 Boehringer Ingelheim Investigational Site, Nottingham
  - 205.235.3616 Boehringer Ingelheim Investigational Site, Paisley
  - 205.235.3614 Boehringer Ingelheim Investigational Site, Penarth
  - 205.235.3603 Boehringer Ingelheim Investigational Site, Plymouth
  - 205.235.3609 Boehringer Ingelheim Investigational Site, Sheffield
  - 205.235.3601 Boehringer Ingelheim Investigational Site, Solihull, Birmingham

REFERENCES:
- [Derived] Rabe KF, Halpin DMG, Han MK, Miravitlles M, Singh D, Gronke L, Voss F, Martinez FJ. Composite endpoints in COPD: clinically important deterioration in the UPLIFT trial. Respir Res. 2020 Jul 9;21(1):177. doi: 10.1186/s12931-020-01431-y. PMID 32646424
- [Derived] Tashkin DP, Miravitlles M, Celli BR, Metzdorf N, Mueller A, Halpin DMG, Anzueto A. Concomitant inhaled corticosteroid use and the risk of pneumonia in COPD: a matched-subgroup post hoc analysis of the UPLIFT(R) trial. Respir Res. 2018 Oct 5;19(1):196. doi: 10.1186/s12931-018-0874-0. PMID 30290801
- [Derived] Celli BR, Decramer M, Liu D, Metzdorf N, Asijee GM, Tashkin DP. Defining a COPD composite safety endpoint for demonstrating efficacy in clinical trials: results from the randomized, placebo-controlled UPLIFT(R) trial. Respir Res. 2016 May 4;17(1):48. doi: 10.1186/s12931-016-0361-4. PMID 27141828
- [Derived] Goossens LM, Leimer I, Metzdorf N, Becker K, Rutten-van Molken MP. Does the 2013 GOLD classification improve the ability to predict lung function decline, exacerbations and mortality: a post-hoc analysis of the 4-year UPLIFT trial. BMC Pulm Med. 2014 Oct 18;14:163. doi: 10.1186/1471-2466-14-163. PMID 25326750
- [Derived] Tashkin DP, Li N, Kleerup EC, Halpin D, Celli B, Decramer M, Elashoff R. Acute bronchodilator responses decline progressively over 4 years in patients with moderate to very severe COPD. Respir Res. 2014 Aug 31;15(1):102. doi: 10.1186/s12931-014-0102-5. PMID 25175805
- [Derived] Janssens W, Liu Y, Liu D, Kesten S, Tashkin DP, Celli BR, Decramer M. Quality and reproducibility of spirometry in COPD patients in a randomized trial (UPLIFT(R)). Respir Med. 2013 Sep;107(9):1409-16. doi: 10.1016/j.rmed.2013.04.015. Epub 2013 May 25. PMID 23714653
- [Derived] Tashkin DP, Celli BR, Decramer M, Lystig T, Liu D, Kesten S. Efficacy of tiotropium in COPD patients with FEV1 >/= 60% participating in the UPLIFT(R) trial. COPD. 2012 Jun;9(3):289-96. doi: 10.3109/15412555.2012.656211. Epub 2012 Mar 20. PMID 22432932
- [Derived] Kesten S, Celli B, Decramer M, Liu D, Tashkin D. Adverse health consequences in COPD patients with rapid decline in FEV1--evidence from the UPLIFT trial. Respir Res. 2011 Sep 28;12(1):129. doi: 10.1186/1465-9921-12-129. PMID 21955733
- [Derived] Tashkin D, Celli B, Kesten S, Lystig T, Decramer M. Effect of tiotropium in men and women with COPD: results of the 4-year UPLIFT trial. Respir Med. 2010 Oct;104(10):1495-504. doi: 10.1016/j.rmed.2010.03.033. Epub 2010 Apr 24. PMID 20418083
- [Derived] Troosters T, Celli B, Lystig T, Kesten S, Mehra S, Tashkin DP, Decramer M; Uplift Investigators. Tiotropium as a first maintenance drug in COPD: secondary analysis of the UPLIFT trial. Eur Respir J. 2010 Jul;36(1):65-73. doi: 10.1183/09031936.00127809. Epub 2010 Feb 25. PMID 20185426
- [Derived] Decramer M, Celli B, Kesten S, Lystig T, Mehra S, Tashkin DP; UPLIFT investigators. Effect of tiotropium on outcomes in patients with moderate chronic obstructive pulmonary disease (UPLIFT): a prespecified subgroup analysis of a randomised controlled trial. Lancet. 2009 Oct 3;374(9696):1171-8. doi: 10.1016/S0140-6736(09)61298-8. Epub 2009 Aug 27. PMID 19716598
- [Derived] Tashkin DP, Celli B, Senn S, Burkhart D, Kesten S, Menjoge S, Decramer M; UPLIFT Study Investigators. A 4-year trial of tiotropium in chronic obstructive pulmonary disease. N Engl J Med. 2008 Oct 9;359(15):1543-54. doi: 10.1056/NEJMoa0805800. Epub 2008 Oct 5. PMID 18836213

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 09 Jan 2003 - 22 Feb 2008; 490 centers in 37 countries
Groups:
- Placebo; Tiotropium Bromide Inhalation Capsules 18 mcg: once daily
Period: Overall Study
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Started | 3006 | 2986
Completed | 1648 | 1887
Not Completed | 1358 | 1099
Not completed — Adverse Event | 746 | 627
Not completed — Protocol Violation | 75 | 48
Not completed — Withdrawal by Subject | 403 | 300
Not completed — Lost to Follow-up | 76 | 64
Not completed — Other | 58 | 60

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg | Total
Number analyzed (Participants) | 3006 | 2986 | 5992
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.52 (8.48) | 64.50 (8.41) | 64.51 (8.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 784 | 735 | 1519.0
  Male | 2222 | 2251 | 4473.0

OUTCOME MEASURES:

1. Primary Outcome: Pre-bronchodilator Forced Expiratory Volume in One Second (FEV1) Rate of Decline From Day 30 to 4 Years
Description: Rate of decline of forced expiratory volume in one second (FEV1) measured before the use of bronchodilators. A negative rate of decline indicates decreasing FEV1 over time, while a positive value indicates increasing FEV1.
Time Frame: From day 30 to 4 years
Measure: Mean (Standard Error); unit: ml/year
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2413 | 2557
ml/year | -30 (1) | -30 (1)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Linear random effects model; Test type: Superiority or Other; p = 0.9524, t-test, 2 sided; Random-effects model; Mean Difference (Final Values) = 0, 95% CI [-4 to 4], Standard Error of Mean 2 — Arbitrary covariance matrix; fixed treatment effect; individual patients are random; rate of decline estimated as the slope of the random effects model

2. Primary Outcome: Post-bronchodilator Forced Expiratory Volume in One Second (FEV1) Rate of Decline From Day 30 to 4 Years
Description: Rate of decline of forced expiratory volume in one second (FEV1) measured after bronchodilation. A negative rate of decline indicates decreasing FEV1 over time, while a positive value indicates increasing FEV1.
Time Frame: From day 30 to 4 years
Measure: Mean (Standard Error); unit: ml/year
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2410 | 2554
ml/year | -42 (1) | -40 (1)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Linear random effects model; Test type: Superiority or Other; p = 0.2074, t-test, 2 sided; Random-effects model; Mean Difference (Final Values) = 2, 95% CI [-2 to 6], Standard Error of Mean 2 — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Pre-bronchodilator Forced Expiratory Volume in One Second (FEV1) Rate of Decline From Day 1 to 30 Days After Completion of Double Blinded Treatment
Description: as for outcome 1
Time Frame: Day 1 to 30 days after completion of double blinded treatment between Day 1 and 4 years plus 30 days.
Measure: Median (Standard Error); unit: ml/year
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 1618 | 1803
ml/year | -17 (2) | -15 (2)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p = 0.2488, Wilcoxon Rank-sum test; Rate calculated as (measure on 30days after completion of treatment - measure on day 1 )/ years in between

4. Secondary Outcome: Post-bronchodilator Forced Expiratory Volume in One Second (FEV1) Rate of Decline From Day 1 to 30 Days After Completion of Double Blinded Treatment
Description: Rate of decline of forced expiratory volume in one second (FEV1) measured after the use of bronchodilators. A negative rate of decline indicates decreasing FEV1 over time, while a positive value indicates increasing FEV1
Time Frame: Day 1 to 30 days after completion of double blinded treatment between Day 1 and 4 years plus 30 days
Measure: Median (Standard Error); unit: ml/year
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 1613 | 1805
ml/year | -32 (2) | -27 (2)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p = 0.0145, Wilcoxon Rank-sum test; Rate calculated as (measure on 30days after completion of treatment - measure on day 1 )/ years in between

5. Secondary Outcome: Pre-bronchodilator Forced Vital Capacity (FVC) Rate of Decline From Day 30 to 4 Years
Description: Rate of decline of forced vital capacity (FVC) measured before the use of bronchodilators. A negative rate of decline indicates decreasing FVC over time, while a positive value indicates increasing FVC
Time Frame: From day 30 to 4 years
Measure: Mean (Standard Error); unit: ml/year
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2413 | 2557
ml/year | -39 (3) | -43 (3)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Linear random effects model; Test type: Superiority or Other; p = 0.2990, t-test, 2 sided; Mean Difference (Final Values) = -4, 95% CI [-12 to 4], Standard Error of Mean 4 — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Post-bronchodilator Forced Vital Capacity (FVC) Rate of Decline From Day 30 to 4 Years
Description: Rate of decline of forced vital capacity (FVC) measured after bronchodilation. A negative rate of decline indicates decreasing FVC over time, while a positive value indicates increasing FVC
Time Frame: From day 30 to 4 years
Measure: Mean (Standard Error); unit: ml/year
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2410 | 2554
ml/year | -61 (3) | -61 (3)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Linear random effects model; Test type: Superiority or Other; p = 0.8375, t-test, 2 sided; Mean Difference (Final Values) = -1, 95% CI [-9 to 7], Standard Error of Mean 4 — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Pre-bronchodilator Slow Vital Capacity (SVC) Rate of Decline From Day 30 to 4 Years
Description: Rate of decline of slow vital capacity (SVC) measured before the use of bronchodilators. A negative rate of decline indicates decreasing SVC over time, while a positive value indicates increasing SVC
Time Frame: From day 30 to 4 years
Measure: Mean (Standard Error); unit: ml/year
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2374 | 2531
ml/year | -41 (3) | -47 (3)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Linear random effects model; Test type: Superiority or Other; p = 0.1143, t-test, 2 sided; Median Difference (Final Values) = -6, 95% CI [-14 to 2], Standard Error of Mean 4 — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Post-bronchodilator Slow Vital Capacity (SVC) Rate of Decline From Day 30 to 4 Years
Description: Rate of decline of slow vital capacity (SVC) measured after bronchodilation. A negative rate of decline indicates decreasing SVC over time, while a positive value indicates increasing SVC
Time Frame: From day 30 to 4 years
Measure: Mean (Standard Error); unit: ml/year
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2383 | 2527
ml/year | -65 (3) | -66 (3)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Linear random effects model; Test type: Superiority or Other; p = 0.7870, t-test, 2 sided; Median Difference (Final Values) = -1, 95% CI [-9 to 7], Standard Error of Mean 4 — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Rate of Decline of St George's Respiratory Questionnaire (SGRQ) Total Score
Description: SGRQ total score shows the impact of COPD on patient's health status, and expressed as a percentage of impairment with scale from 0 (best health status) to 100 (worst possible status). A negative rate of decline shows decreasing SGRQ total score (or improved health) over time, while a positive value shows increasing score (or worsen health).
Time Frame: From month 6 to 4 years
Measure: Mean (Standard Error); unit: Score on scale per year
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2362 | 2505
Score on scale per year | 1.21 (0.09) | 1.25 (0.09)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Linear random effects model; Test type: Superiority or Other; p = 0.7840, t-test, 2 sided; Mean Difference (Final Values) = 0.04, 95% CI [-0.2 to 0.3], Standard Error of Mean 0.13 — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: Pre-bronchodilator Forced Vital Capacity (FVC) Rate of Decline From Day 1 to 30 Days After Completion of Double Blinded Treatment
Description: Rate of decline of forced vital capacity (FVC) before bronchodilation. A negative rate of decline indicates decreasing FVC over time, while a positive value indicates increasing FVC
Time Frame: Day 1 to 30 days after completion of double blinded treatment between Day 1 and 4 years plus 30 days.
Measure: Median (Standard Error); unit: ml/year
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 1618 | 1803
ml/year | -12 (4) | -10 (3)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p = 0.2705, Wilcoxon Rank-sum test; Rate calculated as (measure on 30days after completion of treatment - measure on day 1 )/ years in between

11. Secondary Outcome: Post-bronchodilator Forced Vital Capacity (FVC) Rate of Decline From Day 1 to 30 Days After Completion of Double Blinded Treatment
Description: Rate of decline of forced vital capacity (FVC) after bronchodilation. A negative rate of decline indicates decreasing FVC over time, while a positive value indicates increasing FVC
Time Frame: Day 1 to 30 days after completion of double blinded treatment between Day 1 and 4 years plus 30 days
Measure: Median (Standard Error); unit: ml/year
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 1613 | 1805
ml/year | -40 (4) | -40 (3)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p = 0.306, Wilcoxon Rank-sum test; Rate calculated as (measure on 30days after completion of treatment - measure on day 1 )/ years in between

12. Secondary Outcome: Pre-bronchodilator Slow Vital Capacity (SVC) Rate of Decline From Day 1 to 30 Days After Completion of Double Blinded Treatment
Description: Rate of decline slow vital capacity (SVC) before bronchodilation. A negative rate of decline indicates decreasing SVC over time, while a positive value indicates increasing SVC
Time Frame: Day 1 to 30 days after completion of double blinded treatment between Day 1 and 4 years plus 30 days
Measure: Median (Standard Error); unit: ml/year
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 1562 | 1706
ml/year | -17 (4) | -17 (4)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p = 0.8103, Wilcoxon Rank-sum test; Rate calculated as (measure on 30days after completion of treatment - measure on day 1 )/ years in between

13. Secondary Outcome: Post-bronchodilator Slow Vital Capacity (SVC) Rate of Decline From Day 1 to 30 Days After Completion of Double Blinded Treatment
Description: Rate of decline of slow vital capacity (SVC) after bronchodilation. A negative rate of decline indicates decreasing SVC over time, while a positive value indicates increasing SVC
Time Frame: Day 1 to 30 days after completion of double blinded treatment between Day 1 and 4 years plus 30 days
Measure: Median (Standard Error); unit: ml/year
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 1540 | 1711
ml/year | -46 (4) | -42 (3)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p = 0.9814, Wilcoxon Rank-sum test; Rate calculated as (measure on 30days after completion of treatment - measure on day 1 )/ years in between

14. Secondary Outcome: Time to First Exacerbation
Description: Chronic obstructive pulmonary disease (COPD) exacerbation
Time Frame: From Day 1 to 4 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 3006 | 2986
months | 12.51 [11.53 to 13.79] | 16.65 [14.88 to 17.87]
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Cox regression; Test type: Superiority or Other; p < 0.0001, Log Rank; Cox regression with treatment; Hazard Ratio (HR) = 0.86, 95% CI [0.81 to 0.91], Standard Error of Mean 0.03 — Median estimated by Kaplan-Meier estimates; hazard ratio shown as tio vs. placebo

15. Secondary Outcome: Number of Chronic Obstructive Pulmonary Disease (COPD) Exacerbations Per Patient Year
Time Frame: Day 1 to 4 years
Measure: Mean (Standard Error); unit: number per patient year
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 3006 | 2986
number per patient year | 0.85 (0.02) | 0.73 (0.02)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Poisson regression adjusted for overdispersion and treatment exposure; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Rate Ratio = 0.86, 95% CI [0.81 to 0.91], Standard Error of Mean 0.03 — Ratio calculated as estimated number of events in tio/number of events in placebo

16. Secondary Outcome: Number and Percentage of Patients With at Least One Chronic Obstructive Pulmonary Disease (COPD) Exacerbation
Time Frame: Day 1 to 4 years
Measure: Number; unit: Participants
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 3006 | 2986
Participants
  Number of patients | 2049 | 2001
  Percentage of patients | 68.2 | 67
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p = 0.3481, Fisher Exact

17. Secondary Outcome: Number of Exacerbation Days Per Patient Year
Description: Number of exacerbation days normalized by treatment exposure
Time Frame: Day 1 to 4 years
Measure: Mean (Standard Error); unit: days/patient year
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 3006 | 2986
days/patient year | 13.64 (0.35) | 12.11 (0.32)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Poisson regression adjusted for overdispersion and treatment exposure; Test type: Superiority or Other; p = 0.0011, t-test, 2 sided; Rate Ratio = 0.89, 95% CI [0.83 to 0.95], Standard Error of Mean 0.03 — Poisson regression adjusting for overdispersion with Pearson's method adjusting for treatment exposure. The logarithm of treatment exposure is used as offset when building the Poisson model

18. Secondary Outcome: Time to First COPD Exacerbation Leading to Hospitalization (for 25% Patients)
Time Frame: Day 1 to 4 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 3006 | 2986
months | 28.64 [26.08 to 31.82] | 35.89 [23.38 to 39.54]
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p = 0.1766, Fisher Exact

19. Secondary Outcome: Number and Percentage of Patients With at Least on COPD Exacerbation Leading to Hospitalization
Time Frame: From Day 1 to 4 years
Measure: Number; unit: Participants
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 3006 | 2986
Participants
  Number of patients | 811 | 759
  Percentage of patients | 27 | 25.4
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Cox regression; Test type: Superiority or Other; p = 0.0024, Log Rank; Hazard Ratio (HR) = 0.86, 95% CI [0.78 to 0.95], Standard Error of Mean 0.04 — Hazard ratio shown as tiotropium bromide vs. placebo

20. Secondary Outcome: Number of Exacerbation Leading to Hospitalization
Description: Estimated number of exacerbations leading to hospitalizations per patient year
Time Frame: From Day 1 to 4 years
Measure: Number; unit: Number per patient year
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 3006 | 2986
Number per patient year | 0.16 | 0.15
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p = 0.3413, t-test, 2 sided; Rate ratio = 0.94, 95% CI [0.82 to 1.07], Standard Error of Mean 0.06 — Ratio of estimated number of events between tiotropium bromide and placebo

21. Secondary Outcome: Days of Chronic Obstructive Pulmonary Disease (COPD) Exacerbation Leading to Hospitalization
Description: Number of days with chronic obstructive pulmonary disease (COPD) exacerbation leading to hospitalization (normalized by treatment exposure)
Time Frame: From Day 1 to 4 years
Measure: Mean (Standard Error); unit: days/patient year
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 3006 | 2986
days/patient year | 3.13 (0.17) | 3.17 (0.17)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Poisson regression adjusting for overdispersion with Pearson's method adjusting for treatment exposure. The logarithm of treatment exposure is used as offset when building the Poisson model; Test type: Superiority or Other; p = 0.8624, t-test, 2 sided; Rate ratio = 1.01, 95% CI [0.87 to 1.18] — Ratio of estimated number of days of chronic obstructive pulmonary disease (COPD) exacerbation leading to hospitalization between tio and placebo

22. Secondary Outcome: Estimated Pre-bronchodilator Forced Expiratory Volume in One Second (FEV1) at Month 1
Description: Estimated FEV1 before bronchodilator at Month 1
Time Frame: Month 1
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2363 | 2494
L | 1.134 (0.004) | 1.221 (0.004)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p < .0001, ANOVA; Repeated measures ANOVA; Mean Difference (Final Values) = 0.087, 95% CI [0.077 to 0.098]

23. Secondary Outcome: Estimated Post-bronchodilator Forced Expiratory Volume in One Second (FEV1) at Month 1
Description: Estimated forced expiratory volume in one second (FEV1) after bronchodilator at month 1
Time Frame: Month 1
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2374 | 2516
L | 1.372 (0.004) | 1.418 (0.004)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p < .0001, ANOVA; Repeated measures ANOVA; Mean Difference (Final Values) = 0.047, 95% CI [0.037 to 0.057]

24. Secondary Outcome: Estimated Pre-bronchodilator Forced Expiratory Volume in One Second (FEV1) at Month 6
Description: Estimated forced expiratory volume in one second (FEV1) before bronchodilator at month 6
Time Frame: Month 6
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2363 | 2494
L | 1.126 (0.004) | 1.225 (0.004)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p < .0001, ANOVA; Repeated measures ANOVA; Mean Difference (Final Values) = 0.099, 95% CI [0.087 to 0.110]

25. Secondary Outcome: Estimated Post-bronchodilator Forced Expiratory Volume in One Second (FEV1) at Month 6
Time Frame: Month 6
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2374 | 2516
L | 1.365 (0.004) | 1.423 (0.004)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p < .0001, ANOVA; Repeated measures ANOVA; Mean Difference (Final Values) = 0.058, 95% CI [0.047 to 0.069]

26. Secondary Outcome: Estimated Pre-bronchodilator Forced Expiratory Volume in One Second (FEV1) at Month 12
Time Frame: Month 12
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2363 | 2494
L | 1.111 (0.004) | 1.213 (0.004)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p < .0001, ANOVA; Repeated measures ANOVA; Mean Difference (Final Values) = 0.103, 95% CI [0.091 to 0.115]

27. Secondary Outcome: Estimated Post-bronchodilator Forced Expiratory Volume in One Second (FEV1) at Month 12
Time Frame: Month 12
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2374 | 2516
L | 1.345 (0.004) | 1.398 (0.004)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p < .0001, ANOVA; Repeated measures ANOVA; Median Difference (Final Values) = 0.054, 95% CI [0.042 to 0.065]

28. Secondary Outcome: Estimated Pre-bronchodilator Forced Expiratory Volume in One Second (FEV1) at Month 18
Time Frame: Month 18
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2363 | 2494
L | 1.101 (0.005) | 1.192 (0.005)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p < .0001, ANOVA; Repeated measures ANOVA; Mean Difference (Final Values) = 0.091, 95% CI [0.078 to 0.104]

29. Secondary Outcome: Estimated Post-bronchodilator Forced Expiratory Volume in One Second (FEV1) at Month 18
Time Frame: Month 18
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2374 | 2516
L | 1.326 (0.005) | 1.379 (0.005)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p < .0001, ANOVA; Repeated measures ANOVA; Mean Difference (Final Values) = 0.053, 95% CI [0.040 to 0.066]

30. Secondary Outcome: Estimated Pre-bronchodilator Forced Expiratory Volume in One Second (FEV1) at Month 24
Time Frame: Month 24
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2363 | 2494
L | 1.079 (0.005) | 1.173 (0.005)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p < .0001, ANOVA; Repeated measures ANOVA; Mean Difference (Final Values) = 0.094, 95% CI [0.081 to 0.107]

31. Secondary Outcome: Estimated Post-bronchodilator Forced Expiratory Volume in One Second (FEV1) at Month 24
Time Frame: Month 24
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2374 | 2516
L | 1.294 (0.005) | 1.356 (0.005)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p < .0001, ANOVA; Repeated measures ANOVA; Mean Difference (Final Values) = 0.062, 95% CI [0.049 to 0.075]

32. Secondary Outcome: Estimated Pre-bronchodilator Forced Expiratory Volume in One Second (FEV1) at Month 30
Time Frame: Month 30
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2363 | 2494
L | 1.061 (0.005) | 1.156 (0.005)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p < .0001, ANOVA; Repeated measures ANOVA; Mean Difference (Final Values) = 0.095, 95% CI [0.081 to 0.109]

33. Secondary Outcome: Estimated Post-bronchodilator Forced Expiratory Volume in One Second (FEV1) at Month 30
Time Frame: Month 30
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2374 | 2516
L | 1.274 (0.005) | 1.335 (0.005)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p < .0001, ANOVA; Repeated measures ANOVA; Mean Difference (Final Values) = 0.061, 95% CI [0.047 to 0.075]

34. Secondary Outcome: Estimated Pre-bronchodilator Forced Expiratory Volume in One Second (FEV1) at Month 36
Time Frame: Month 36
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2363 | 2494
L | 1.045 (0.005) | 1.144 (0.005)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p < .0001, ANOVA; Repeated measures ANOVA; Mean Difference (Final Values) = 0.099, 95% CI [0.085 to 0.114]

35. Secondary Outcome: Estimated Post-bronchodilator Forced Expiratory Volume in One Second (FEV1) at Month 36
Time Frame: Month 36
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2374 | 2516
L | 1.250 (0.005) | 1.315 (0.005)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p < .0001, ANOVA; Repeated measures ANOVA; Mean Difference (Final Values) = 0.065, 95% CI [0.051 to 0.080]

36. Secondary Outcome: Estimated Pre-bronchodilator Forced Expiratory Volume in One Second (FEV1) at Month 42
Time Frame: Month 42
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2363 | 2494
L | 1.034 (0.005) | 1.129 (0.005)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p < .0001, ANOVA; Repeated measures ANOVA; Mean Difference (Final Values) = 0.095, 95% CI [0.080 to 0.110]

37. Secondary Outcome: Estimated Post-bronchodilator Forced Expiratory Volume in One Second (FEV1) at Month 42
Description: Estimated FEV1 after bronchodilator at Month 42
Time Frame: Month 42
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2374 | 2516
L | 1.236 (0.006) | 1.297 (0.005)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p < .0001, ANOVA; Repeated measures ANOVA; Mean Difference (Final Values) = 0.061, 95% CI [0.045 to 0.076]

38. Secondary Outcome: Estimated Pre-bronchodilator Forced Expiratory Volume in One Second (FEV1) at Month 48
Time Frame: Month 48
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2363 | 2494
L | 1.024 (0.006) | 1.112 (0.005)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p < .0001, ANOVA; Repeated measures ANOVA; Mean Difference (Final Values) = 0.088, 95% CI [0.073 to 0.103]

39. Secondary Outcome: Estimated Post-bronchodilator Forced Expiratory Volume in One Second (FEV1) at Month 48
Time Frame: Month 48
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2374 | 2516
L | 1.219 (0.006) | 1.268 (0.006)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p < .0001, ANOVA; Repeated measures ANOVA; Mean Difference (Final Values) = 0.049, 95% CI [0.033 to 0.065]

40. Secondary Outcome: Estimated Pre-bronchodilator Forced Vital Capacity (FVC) at Month 1
Time Frame: Month 1
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2363 | 2494
L | 2.667 (0.008) | 2.856 (0.008)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p < .0001, ANOVA; Repeated measures ANOVA; Mean Difference (Final Values) = 0.190, 95% CI [0.168 to 0.211]

41. Secondary Outcome: Estimated Post-bronchodilator Forced Vital Capacity (FVC) at Month 1
Time Frame: Month 1
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2374 | 2516
L | 3.149 (0.007) | 3.204 (0.006)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p < .0001, ANOVA; Repeated measures ANOVA; Mean Difference (Final Values) = 0.055, 95% CI [0.037 to 0.073]

42. Secondary Outcome: Estimated Pre-bronchodilator Forced Vital Capacity (FVC) at Month 6
Time Frame: Month 6
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2363 | 2494
L | 2.658 (0.009) | 2.862 (0.008)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p < .0001, ANOVA; Repeated measures ANOVA; Mean Difference (Final Values) = 0.204, 95% CI [0.180 to 0.228]

43. Secondary Outcome: Estimated Post-bronchodilator Forced Vital Capacity (FVC) at Month 6
Time Frame: Month 6
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2374 | 2516
L | 3.137 (0.008) | 3.193 (0.007)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p < .0001, ANOVA; Repeated measures ANOVA; Mean Difference (Final Values) = 0.055, 95% CI [0.034 to 0.076]

44. Secondary Outcome: Estimated Pre-bronchodilator Forced Vital Capacity (FVC) at Month 12
Time Frame: Month 12
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2363 | 2494
L | 2.640 (0.009) | 2.838 (0.009)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p < .0001, ANOVA; Repeated measures ANOVA; Mean Difference (Final Values) = 0.198, 95% CI [0.173 to 0.222]

45. Secondary Outcome: Estimated Post-bronchodilator Forced Vital Capacity (FVC) at Month 12
Time Frame: Month 12
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2374 | 2516
L | 3.110 (0.008) | 3.158 (0.008)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p < .0001, ANOVA; Repeated measures ANOVA; Mean Difference (Final Values) = 0.048, 95% CI [0.026 to 0.070]

46. Secondary Outcome: Estimated Pre-bronchodilator Forced Vital Capacity (FVC) at Month 18
Time Frame: Month 18
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2363 | 2494
L | 2.622 (0.010) | 2.816 (0.010)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p < .0001, ANOVA; Repeated measures ANOVA; Mean Difference (Final Values) = 0.194, 95% CI [0.167 to 0.221]

47. Secondary Outcome: Estimated Post-bronchodilator Forced Vital Capacity (FVC) at Month 18
Time Frame: Month 18
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2374 | 2516
L | 3.075 (0.009) | 3.126 (0.009)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p < .0001, ANOVA; Repeated measures ANOVA; Mean Difference (Final Values) = 0.050, 95% CI [0.026 to 0.074]

48. Secondary Outcome: Estimated Pre-bronchodilator Forced Vital Capacity (FVC) at Month 24
Time Frame: Month 24
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2363 | 2494
L | 2.597 (0.010) | 2.785 (0.010)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p < .0001, ANOVA; Repeated measures ANOVA; Mean Difference (Final Values) = 0.189, 95% CI [0.161 to 0.216]

49. Secondary Outcome: Estimated Post-bronchodilator Forced Vital Capacity (FVC) at Month 24
Time Frame: Month 24
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2374 | 2516
L | 3.036 (0.009) | 3.095 (0.009)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p < .0001, ANOVA; Repeated measures ANOVA; Mean Difference (Final Values) = 0.059, 95% CI [0.035 to 0.084]

50. Secondary Outcome: Estimated Pre-bronchodilator Forced Vital Capacity (FVC) at Month 30
Time Frame: Month 30
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2363 | 2494
L | 2.572 (0.010) | 2.757 (0.010)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p < .0001, ANOVA; Repeated measures ANOVA; Mean Difference (Final Values) = 0.185, 95% CI [0.157 to 0.213]

51. Secondary Outcome: Estimated Post-bronchodilator Forced Vital Capacity (FVC) at Month 30
Time Frame: Month 30
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2374 | 2516
L | 3.010 (0.010) | 3.057 (0.009)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p = 0.0005, ANOVA; Repeated measures ANOVA; Mean Difference (Final Values) = 0.047, 95% CI [0.021 to 0.074]

52. Secondary Outcome: Estimated Pre-bronchodilator Forced Vital Capacity (FVC) at Month 36
Time Frame: Month 36
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2363 | 2494
L | 2.553 (0.011) | 2.753 (0.010)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p < .0001, ANOVA; Repeated measures ANOVA; Mean Difference (Final Values) = 0.200, 95% CI [0.170 to 0.229]

53. Secondary Outcome: Estimated Post-bronchodilator Forced Vital Capacity (FVC) at Month 36
Time Frame: Month 36
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2374 | 2516
L | 2.973 (0.010) | 3.038 (0.010)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p < .0001, ANOVA; Repeated measures ANOVA; Mean Difference (Final Values) = 0.065, 95% CI [0.038 to 0.093]

54. Secondary Outcome: Estimated Pre-bronchodilator Forced Vital Capacity (FVC) at Month 42
Time Frame: Month 42
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2363 | 2494
L | 2.540 (0.011) | 2.724 (0.011)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p < .0001, ANOVA; Repeated measures ANOVA; Mean Difference (Final Values) = 0.184, 95% CI [0.154 to 0.215]

55. Secondary Outcome: Estimated Post-bronchodilator Forced Vital Capacity (FVC) at Month 42
Time Frame: Month 42
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2374 | 2516
L | 2.959 (0.011) | 3.005 (0.010)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p = 0.0020, ANOVA; Repeated measures ANOVA; Mean Difference (Final Values) = 0.046, 95% CI [0.017 to 0.076]

56. Secondary Outcome: Estimated Pre-bronchodilator Forced Vital Capacity (FVC) at Month 48
Time Frame: Month 48
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2363 | 2494
L | 2.532 (0.011) | 2.702 (0.011)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p < .0001, ANOVA; Repeated measures ANOVA; Mean Difference (Final Values) = 0.170, 95% CI [0.139 to 0.201]

57. Secondary Outcome: Estimated Post-bronchodilator Forced Vital Capacity (FVC) at Month 48
Time Frame: Month 48
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2374 | 2516
L | 2.929 (0.011) | 2.961 (0.010)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p = 0.0365, ANOVA; Repeated measures ANOVA; Mean Difference (Final Values) = 0.032, 95% CI [0.002 to 0.061]

58. Secondary Outcome: Estimated Pre-bronchodilator Slow Vital Capacity (SVC) at Month 1
Time Frame: Month 1
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2325 | 2447
L | 2.847 (0.008) | 3.017 (0.008)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p < .0001, ANOVA; Repeated measures ANOVA; Mean Difference (Final Values) = 0.170, 95% CI [0.147 to 0.192]

59. Secondary Outcome: Estimated Post-bronchodilator Slow Vital Capacity (SVC) at Month 1
Time Frame: Month 1
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2340 | 2467
L | 3.280 (0.007) | 3.318 (0.007)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p = 0.0002, ANOVA; Repeated measures ANOVA; Mean Difference (Final Values) = 0.038, 95% CI [0.018 to 0.058]

60. Secondary Outcome: Estimated Pre-bronchodilator Slow Vital Capacity (SVC) at Month 6
Time Frame: Month 6
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2325 | 2447
L | 2.841 (0.009) | 3.027 (0.009)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p < .0001, ANOVA; Repeated measures ANOVA; Mean Difference (Final Values) = 0.186, 95% CI [0.161 to 0.210]

61. Secondary Outcome: Estimated Post-bronchodilator Slow Vital Capacity (SVC) at Month 6
Time Frame: Month 6
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2340 | 2467
L | 3.268 (0.008) | 3.304 (0.008)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p = 0.0018, ANOVA; Repeated measures ANOVA; Mean Difference (Final Values) = 0.037, 95% CI [0.014 to 0.060]

62. Secondary Outcome: Estimated Pre-bronchodilator Slow Vital Capacity (SVC) at Month 12
Time Frame: Month 12
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2325 | 2447
L | 2.820 (0.009) | 2.996 (0.009)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p < .0001, ANOVA; Repeated measures ANOVA; Mean Difference (Final Values) = 0.176, 95% CI [0.151 to 0.201]

63. Secondary Outcome: Estimated Post-bronchodilator Slow Vital Capacity (SVC) at Month 12
Time Frame: Month 12
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2340 | 2467
L | 3.228 (0.008) | 3.260 (0.008)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p = 0.0069, ANOVA; Repeated measures ANOVA; Mean Difference (Final Values) = 0.032, 95% CI [0.009 to 0.055]

64. Secondary Outcome: Estimated Pre-bronchodilator Slow Vital Capacity (SVC) at Month 18
Time Frame: Month 18
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2325 | 2447
L | 2.811 (0.010) | 2.965 (0.010)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p < .0001, ANOVA; Repeated measures ANOVA; Mean Difference (Final Values) = 0.154, 95% CI [0.127 to 0.182]

65. Secondary Outcome: Estimated Post-bronchodilator Slow Vital Capacity (SVC) at Month 18
Time Frame: Month 18
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2340 | 2467
L | 3.195 (0.009) | 3.234 (0.009)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p = 0.0020, ANOVA; Repeated measures ANOVA; Mean Difference (Final Values) = 0.040, 95% CI [0.015 to 0.065]

66. Secondary Outcome: Estimated Pre-bronchodilator Slow Vital Capacity (SVC) at Month 24
Time Frame: Month 24
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2325 | 2447
L | 2.775 (0.010) | 2.942 (0.010)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p < .0001, ANOVA; Repeated measures ANOVA; Mean Difference (Final Values) = 0.167, 95% CI [0.139 to 0.194]

67. Secondary Outcome: Estimated Post-bronchodilator Slow Vital Capacity (SVC) at Month 24
Time Frame: Month 24
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2340 | 2467
L | 3.157 (0.009) | 3.189 (0.009)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p = 0.0165, ANOVA; Repeated measures ANOVA; Mean Difference (Final Values) = 0.032, 95% CI [0.006 to 0.057]

68. Secondary Outcome: Estimated Pre-bronchodilator Slow Vital Capacity (SVC) at Month 30
Time Frame: Month 30
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2325 | 2447
L | 2.738 (0.011) | 2.908 (0.010)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p < .0001, ANOVA; Repeated measures ANOVA; Mean Difference (Final Values) = 0.170, 95% CI [0.141 to 0.199]

69. Secondary Outcome: Estimated Post-bronchodilator Slow Vital Capacity (SVC) at Month 30
Time Frame: Month 30
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2340 | 2467
L | 3.126 (0.010) | 3.157 (0.010)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p = 0.0248, ANOVA; Repeated measures ANOVA; Mean Difference (Final Values) = 0.031, 95% CI [0.004 to 0.059]

70. Secondary Outcome: Estimated Pre-bronchodilator Slow Vital Capacity (SVC) at Month 36
Time Frame: Month 36
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2325 | 2447
L | 2.731 (0.011) | 2.897 (0.010)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p < .0001, ANOVA; Repeated measures ANOVA; Mean Difference (Final Values) = 0.166, 95% CI [0.136 to 0.196]

71. Secondary Outcome: Estimated Post-bronchodilator Slow Vital Capacity (SVC) at Month 36
Time Frame: Month 36
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2340 | 2467
L | 3.086 (0.010) | 3.136 (0.010)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p = 0.0004, ANOVA; Repeated measures ANOVA; Mean Difference (Final Values) = 0.050, 95% CI [0.022 to 0.078]

72. Secondary Outcome: Estimated Pre-bronchodilator Slow Vital Capacity (SVC) at Month 42
Time Frame: Month 42
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2325 | 2447
L | 2.713 (0.011) | 2.875 (0.011)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p < .0001, ANOVA; Repeated measures ANOVA; Mean Difference (Final Values) = 0.161, 95% CI [0.130 to 0.192]

73. Secondary Outcome: Estimated Post-bronchodilator Slow Vital Capacity (SVC) at Month 42
Time Frame: Month 42
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2340 | 2467
L | 3.073 (0.011) | 3.100 (0.011)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p = 0.0809, ANOVA; Repeated measures ANOVA; Mean Difference (Final Values) = 0.027, 95% CI [-0.003 to 0.057]

74. Secondary Outcome: Estimated Pre-bronchodilator Slow Vital Capacity (SVC) at Month 48
Time Frame: Month 48
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2325 | 2447
L | 2.696 (0.012) | 2.846 (0.011)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p < .0001, ANOVA; Repeated measures ANOVA; Mean Difference (Final Values) = 0.150, 95% CI [0.119 to 0.182]

75. Secondary Outcome: Estimated Post-bronchodilator Slow Vital Capacity (SVC) at Month 48
Time Frame: Month 48
Measure: Mean (Standard Error); unit: L
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2340 | 2467
L | 3.041 (0.011) | 3.067 (0.011)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p = 0.0915, ANOVA; Repeated measures ANOVA; Mean Difference (Final Values) = 0.026, 95% CI [-0.004 to 0.057]

76. Secondary Outcome: Estimated St George's Respiratory Questionnaire (SGRQ) Total Score at Month 6
Description: * SGRQ total score summarizes the impact of COPD on overall patient's health status.
  * Total scores are expressed as a percentage of overall impairment where 100 represents worst possible health status and 0 indicates best possible health status.
  * The scale is continuous.
  * Rate of decline shows the yearly change of SGRQ total score.
Time Frame: Month 6
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2337 | 2478
Units on a scale | 42.289 (0.240) | 39.409 (0.233)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p < .0001, ANOVA; Repeated measures ANOVA; Mean Difference (Final Values) = -2.880, 95% CI [-3.535 to -2.226]

77. Secondary Outcome: Estimated St George's Respiratory Questionnaire (SGRQ) Total Score at Month 12
Description: as for outcome 76
Time Frame: Month 12
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2337 | 2478
Units on a scale | 42.501 (0.253) | 39.730 (0.245)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p < .0001, ANOVA; Repeated measures ANOVA; Mean Difference (Final Values) = -2.771, 95% CI [-3.461 to -2.081]

78. Secondary Outcome: Estimated St George's Respiratory Questionnaire (SGRQ) Total Score at Month 18
Description: as for outcome 76
Time Frame: Month 18
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2337 | 2478
Units on a scale | 43.067 (0.278) | 40.474 (0.269)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p < .0001, ANOVA; Repeated measures ANOVA; Mean Difference (Final Values) = -2.593, 95% CI [-3.352 to -1.834]

79. Secondary Outcome: Estimated St George's Respiratory Questionnaire (SGRQ) Total Score at Month 24
Description: as for outcome 76
Time Frame: Month 24
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2337 | 2478
Units on a scale | 43.562 (0.297) | 41.178 (0.286)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p < .0001, ANOVA; Repeated measures ANOVA; Mean Difference (Final Values) = -2.384, 95% CI [-3.191 to -1.576]

80. Secondary Outcome: Estimated St George's Respiratory Questionnaire (SGRQ) Total Score at Month 30
Description: as for outcome 76
Time Frame: Month 30
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2337 | 2478
Units on a scale | 44.342 (0.315) | 41.919 (0.301)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p < .0001, ANOVA; Repeated measures ANOVA; Mean Difference (Final Values) = -2.423, 95% CI [-3.277 to -1.569]

81. Secondary Outcome: Estimated St George's Respiratory Questionnaire (SGRQ) Total Score at Month 36
Description: as for outcome 76
Time Frame: Month 36
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2337 | 2478
Units on a scale | 45.280 (0.326) | 41.935 (0.311)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p < .0001, ANOVA; Repeated measures ANOVA; Mean Difference (Final Values) = -3.345, 95% CI [-4.229 to -2.462]

82. Secondary Outcome: Estimated St George's Respiratory Questionnaire (SGRQ) Total Score at Month 42
Description: as for outcome 76
Time Frame: Month 42
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2337 | 2478
Units on a scale | 45.722 (0.342) | 42.905 (0.325)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p < .0001, ANOVA; Repeated measures ANOVA; Mean Difference (Final Values) = -2.818, 95% CI [-3.742 to -1.894]

83. Secondary Outcome: Estimated St George's Respiratory Questionnaire (SGRQ) Total Score at Month 48
Description: as for outcome 76
Time Frame: Month 48
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 2337 | 2478
Units on a scale | 45.968 (0.357) | 43.665 (0.338)
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p < .0001, ANOVA; Repeated measures ANOVA; Mean Difference (Final Values) = -2.303, 95% CI [-3.266 to -1.340]

84. Secondary Outcome: Number and Percentage of Participants With All Cause Death and Time to Event Analysis (On-treatment)
Description: On-treatment defined as day 1 to completion of double blinded treatment plus 30 days
Time Frame: Day 1 to completion of double blinded treatment plus 30 days between Day 1 and 4 years plus 30 days
Measure: Number; unit: Participants
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 3006 | 2986
Participants
  Number of patients with on-treatment death | 402 | 374
  Percentage patients with on-treatment death | 13.4 | 12.5
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p = 0.0242, Log Rank; Hazard Ratio (HR) = 0.85, 95% CI [0.74 to 0.98], Standard Error of Mean 0.06 — Cox regression with treatment; hazard ratio shown as tiotropium bromide vs. placebo

85. Post Hoc Outcome: Number and Percentage of Participants With All Cause Death (Including Vital Status Follow-up, Cutoff at 1440 Days)
Time Frame: Day 1 to day 1440
Measure: Number; unit: Participants
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 3006 | 2986
Participants
  Number of patients died from day 1 to day 1440 | 491 | 430
  Percentage of patients died from day 1 to day 1440 | 16.3 | 14.4
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Hazard ratio of all cause mortality vital status was information followed-up after discontinuation; vital status information up to 1440 days after the start of treatment was used; Test type: Superiority or Other; p = 0.0339, Log Rank; Hazard Ratio (HR) = 0.87, 95% CI [0.76 to 0.99], Standard Error of Mean 0.06 — Cox regression; cut-off at 4 years ; vital status form intended at 4 years; hazard ratio shown as tio vs. placebo

86. Secondary Outcome: Number and Percentage of Participants With All Cause Death (Including Vital Status Follow-up, Cutoff at 1470 Days)
Description: All cause mortality vital status information was followed-up after discontinuation; vital status information up to 1470 days after the start of treatment was used.
Time Frame: Day 1 to day 1470
Measure: Number; unit: Participants
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 3006 | 2986
Participants
  Number of patients died from day 1 to day 1470 | 495 | 446
  Percentage of patients died from day 1 to day 1470 | 16.5 | 14.9
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p = 0.0859, Log Rank; Hazard Ratio (HR) = 0.89, 95% CI [0.79 to 1.02], Standard Error of Mean 0.06 — Cox regression; cut-off at 4 years plus 30 days; vital status form intended at 4 years; hazard ratio shown as tio vs. placebo

87. Secondary Outcome: Number and Percentage of Participants With Lower Respiratory Death (On-treatment; Adjudicated Primary Cause)
Description: The primary cause of death was adjudicated by an external committee prior to unblinding; on-treatment defined as day 1 to completion of double blinded treatment plus 30 days
Time Frame: Day 1 to completion of double blinded treatment plus 30 days between Day 1 and 4 years plus 30 days
Measure: Number; unit: Participants
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 3006 | 2986
Participants
  Number of patients with lower respiratory | 140 | 131
  Percentage of patients with lower respiratory | 4.7 | 4.4
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p = 0.1936, Log Rank; Hazard Ratio (HR) = 0.85, 95% CI [0.67 to 1.08] — Cox regression with treatment; hazard ratio shown as tiotropium bromide vs. placebo

88. Secondary Outcome: Number and Percentage of Participants With a Lower Respiratory Death (Adjudicated; Including Vital Status Follow-up, Cutoff at 1470 Days)
Description: The primary cause of death was adjudicated by an external committee prior to unblinding; vital status was information followed-up after discontinuation; vital status information up to 1470 days after the start of treatment was used
Time Frame: Day 1 to day 1470
Measure: Number; unit: Participants
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 3006 | 2986
Participants
  Number of patients with lower respiratory death | 173 | 153
  Percentage patients with lower respiratory death | 5.8 | 5.1
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p = 0.2377, Log Rank; Hazard Ratio (HR) = 0.88, 95% CI [0.71 to 1.09] — Cox regression; cut-off at 4 years plus 30 days; vital status form intended at 4 years; hazard ratio shown as tiotropium bromide vs. placebo

89. Other Pre Specified Outcome: Incidence Rate of Serious Adverse Event (System Organ Class = Cardiac Disorders)
Description: Descriptive statistics show the number of patients with event, central tendency shows incidence rate. Incidence rate calculated as number of patients with event divided by at-risk years * 100.
Time Frame: Day 1 to completion of double blinded treatment plus 30 days
Measure: Number; unit: Number of patients with event
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 3006 | 2986
Number of patients with event
  Number of patients with event | 350 | 322
  Incidence rate (number of events/100 patient year) | 4.21 | 3.56
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p = 0.0290, Z-test; incidence rate = number of patients with event/ time at risk; Rate ratio of incidence rates = 0.84, 95% CI [0.73 to 0.98] — Rate ratio of incidence rates (tiotropium/placebo)

90. Other Pre Specified Outcome: Incidence Rate of Serious Adverse Event (Preferred Term = Angina)
Description: as for outcome 89
Time Frame: Day 1 to completion of double blinded treatment plus 30 days
Measure: Number; unit: Number of patients with event
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 3006 | 2986
Number of patients with event
  Number of patients with event | 31 | 48
  Incidence rate (number events/100-patient years) | 0.36 | 0.51
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p = 0.1158, Z-test; Rate ratio of incidence rates = 1.44, 95% CI [0.91 to 2.26] — Rate ratio of incidence rates (tiotropium/placebo)

91. Other Pre Specified Outcome: Incidence Rate of Serious Adverse Event (Preferred Term = Atrial Fibrillation)
Description: as for outcome 89
Time Frame: Day 1 to completion of double blinded treatment plus 30 days
Measure: Number; unit: Number of patients with event
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 3006 | 2986
Number of patients with event
  Number of patients with event | 67 | 69
  Incidence rate (number events/100-patient years) | 0.77 | 0.74
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p = 0.7725, Z-test; Rate ratio of incidence rates = 0.95, 95% CI [0.68 to 1.33] — Rate ratio of incidence rates (tiotropium/placebo)

92. Other Pre Specified Outcome: Incidence Rate of Serious Adverse Event (Preferred Term = Cardiac Failure)
Description: as for outcome 89
Time Frame: Day 1 to completion of double blinded treatment plus 30 days
Measure: Number; unit: Number of patients with event
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 3006 | 2986
Number of patients with event
  Number of patients with event | 42 | 57
  Incidence rate (number events/100-patient years) | 0.48 | 0.61
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p = 0.2666, Z-test; Rate ratio of incidence rates = 1.25, 95% CI [0.84 to 1.87] — Rate ratio of incidence rates (tiotropium/placebo)

93. Other Pre Specified Outcome: Incidence Rate of Serious Adverse Event (Preferred Term = Cardiac Failure Congestive)
Description: as for outcome 89
Time Frame: Day 1 to completion of double blinded treatment plus 30 days
Measure: Number; unit: Number of patients with event
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 3006 | 2986
Number of patients with event
  Number of patients with event | 42 | 27
  Incidence rate (number events/100-patient years) | 0.48 | 0.29
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p = 0.0337, Z-test; Rate ratio of incidence rates = 0.59, 95% CI [0.37 to 0.96] — Rate ratio of incidence rates (tiotropium/placebo)

94. Other Pre Specified Outcome: Incidence Rate of Serious Adverse Event (Preferred Term = Coronary Artery Disease)
Description: as for outcome 89
Time Frame: Day 1 to completion of double blinded treatment plus 30 days
Measure: Number; unit: Number of patients with event
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 3006 | 2986
Number of patients with event
  Number of patients with event | 32 | 20
  Incidence rate (number events/100-patient years) | 0.37 | 0.21
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p = 0.0537, Z-test; Rate ratio of incidence rates = 0.58, 95% CI [0.33 to 1.01] — Rate ratio of incidence rates (tiotropium/placebo)

95. Other Pre Specified Outcome: Incidence Rate of Serious Adverse Event (Preferred Term = Myocardial Infarction)
Description: as for outcome 89
Time Frame: Day 1 to completion of double blinded treatment plus 30 days
Measure: Number; unit: Number of patients with event
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 3006 | 2986
Number of patients with event
  Number of patients with event | 84 | 65
  Incidence rate (number events/100-patient years) | 0.97 | 0.69
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p = 0.0403, Z-test; Rate ratio of incidence rates = 0.71, 95% CI [0.52 to 0.99] — Rate ratio of incidence rates (tiotropium/placebo)

96. Other Pre Specified Outcome: Incidence Rate of Serious Adverse Event (System Organ Class = Lower Respiratory System Disorders)
Description: as for outcome 89
Time Frame: Day 1 to completion of double blinded treatment plus 30 days
Measure: Number; unit: Number of patients with event
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 3006 | 2986
Number of patients with event
  Number of patients with event | 985 | 911
  Incidence rate (number events/100-patient years) | 13.47 | 11.32
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p = 0.0001, Z-test; Rate ratio of incidence rates = 0.84, 95% CI [0.77 to 0.92] — Rate ratio of incidence rates (tiotropium/placebo)

97. Other Pre Specified Outcome: Incidence Rate of Serious Adverse Event (Preferred Term = Bronchitis)
Description: as for outcome 89
Time Frame: Day 1 to completion of double blinded treatment plus 30 days
Measure: Number; unit: Number of patients with event
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 3006 | 2986
Number of patients with event
  Number of patients with event | 27 | 35
  Incidence rate (number events/100-patient years) | 0.31 | 0.37
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p = 0.4789, Z-test; Rate ratio of incidence rates = 1.20, 95% CI [0.73 to 1.98] — Rate ratio of incidence rates (tiotropium/placebo)

98. Other Pre Specified Outcome: Incidence Rate of Serious Adverse Event (Preferred Term = Chronic Obstructive Pulmonary Disease (COPD) Exacerbation)
Description: as for outcome 89
Time Frame: Day 1 to completion of double blinded treatment plus 30 days
Measure: Number; unit: Number of patients with event
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 3006 | 2986
Number of patients with event
  Number of patients with event | 742 | 688
  Incidence rate (number events/100-patient years) | 9.70 | 8.19
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p = 0.0014, Z-test; Rate ratio of incidence rates = 0.84, 95% CI [0.76 to 0.94] — Rate ratio of incidence rates (tiotropium/placebo)

99. Other Pre Specified Outcome: Incidence Rate of Serious Adverse Event (Preferred Term = Dyspnoea)
Description: as for outcome 89
Time Frame: Day 1 to completion of double blinded treatment plus 30 days
Measure: Number; unit: Number of patients with event
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 3006 | 2986
Number of patients with event
  Number of patients with event | 54 | 36
  Incidence rate (number events/100-patient years) | 0.62 | 0.38
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p = 0.0236, Z-test; Rate ratio of incidence rates = 0.61, 95% CI [0.40 to 0.94] — Rate ratio of incidence rates (tiotropium/placebo)

100. Other Pre Specified Outcome: Incidence Rate of Serious Adverse Event (Preferred Term = Pneumonia)
Description: as for outcome 89
Time Frame: Day 1 to completion of double blinded treatment plus 30 days
Measure: Number; unit: Number of patients with event
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 3006 | 2986
Number of patients with event
  Number of patients with event | 290 | 296
  Incidence rate (number events/100-patient years) | 3.46 | 3.28
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p = 0.5064, Z-test; Rate ratio of incidence rates = 0.95, 95% CI [0.81 to 1.11] — Rate ratio of incidence rates (tiotropium/placebo)

101. Other Pre Specified Outcome: Incidence Rate of Serious Adverse Event (Preferred Term = Respiratory Failure)
Description: as for outcome 89
Time Frame: Day 1 to completion of double blinded treatment plus 30 days
Measure: Number; unit: Number of patients with event
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Number analyzed (Participants) | 3006 | 2986
Number of patients with event
  Number of patients with event | 113 | 85
  Incidence rate (number events/100-patient years) | 1.31 | 0.90
Statistical Analysis 1: Comparison: Placebo vs Tiotropium Bromide Inhalation Capsules 18 mcg; Test type: Superiority or Other; p = 0.0104, Z-test; Rate ratio of incidence rates = 0.69, 95% CI [0.52 to 0.92] — Rate ratio of incidence rates (tiotropium/placebo)

ADVERSE EVENTS:
Time Frame: From first drug administration until 30 days after last drug administration
Description: The Dictionary used to report the adverse events is Sponsor-defined based on the MedDRA version 11.0
Arm/Group | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Serious Adverse Events (participants affected / at risk) | 1509 | 1540
Other Adverse Events (participants affected / at risk) | 2622 | 2643
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Anaemia (Blood and lymphatic system disorders) | 11/3006 | 19/2986
Coagulopathy (Blood and lymphatic system disorders) | 0/3006 | 2/2986
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1/3006 | 0/2986
Febrile neutropenia (Blood and lymphatic system disorders) | 2/3006 | 1/2986
Haemolytic anaemia (Blood and lymphatic system disorders) | 1/3006 | 0/2986
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 4/3006 | 0/2986
Hypocoagulable state (Blood and lymphatic system disorders) | 0/3006 | 1/2986
Iron deficiency anaemia (Blood and lymphatic system disorders) | 4/3006 | 2/2986
Leukocytosis (Blood and lymphatic system disorders) | 0/3006 | 1/2986
Leukopenia (Blood and lymphatic system disorders) | 0/3006 | 1/2986
Lymphadenopathy (Blood and lymphatic system disorders) | 1/3006 | 0/2986
Microcytic anaemia (Blood and lymphatic system disorders) | 1/3006 | 1/2986
Neutropenia (Blood and lymphatic system disorders) | 0/3006 | 2/2986
Polycythaemia (Blood and lymphatic system disorders) | 1/3006 | 2/2986
Splenic haemorrhage (Blood and lymphatic system disorders) | 0/3006 | 1/2986
Splenic lesion (Blood and lymphatic system disorders) | 0/3006 | 1/2986
Splenic vein thrombosis (Blood and lymphatic system disorders) | 1/3006 | 0/2986
Splenomegaly (Blood and lymphatic system disorders) | 1/3006 | 0/2986
Thrombocytopenia (Blood and lymphatic system disorders) | 3/3006 | 0/2986
Accelerated idioventricular rhythm (Cardiac disorders) | 1/3006 | 0/2986
Acute coronary syndrome (Cardiac disorders) | 2/3006 | 6/2986
Acute right ventricular failure (Cardiac disorders) | 0/3006 | 1/2986
Angina (Cardiac disorders) | 31/3006 | 48/2986
Aortic valve disease (Cardiac disorders) | 1/3006 | 0/2986
Aortic valve incompetence (Cardiac disorders) | 2/3006 | 0/2986
Aortic valve stenosis (Cardiac disorders) | 0/3006 | 2/2986
Arrhythmia (Cardiac disorders) | 10/3006 | 7/2986
Arrhythmia supraventricular (Cardiac disorders) | 1/3006 | 1/2986
Arteriosclerosis coronary artery (Cardiac disorders) | 1/3006 | 1/2986
Atrial Fibrillation (Cardiac disorders) | 67/3006 | 69/2986
Atrial tachycardia (Cardiac disorders) | 0/3006 | 2/2986
Atrial thrombosis (Cardiac disorders) | 1/3006 | 0/2986
Atrioventricular block (Cardiac disorders) | 1/3006 | 3/2986
Atrioventricular block complete (Cardiac disorders) | 4/3006 | 5/2986
Atrioventricular block first degree (Cardiac disorders) | 0/3006 | 1/2986
Atrioventricular block second degree (Cardiac disorders) | 3/3006 | 1/2986
Bradycardia (Cardiac disorders) | 5/3006 | 1/2986
Bundle branch block left (Cardiac disorders) | 0/3006 | 1/2986
Bundle branch block right (Cardiac disorders) | 1/3006 | 0/2986
Cardiac aneurysm (Cardiac disorders) | 1/3006 | 0/2986
Cardiac arrest (Cardiac disorders) | 11/3006 | 6/2986
Cardiac asthma (Cardiac disorders) | 0/3006 | 1/2986
Cardiac disorder (Cardiac disorders) | 2/3006 | 0/2986
Cardiac failure (Cardiac disorders) | 42/3006 | 57/2986
Cardiac failure acute (Cardiac disorders) | 3/3006 | 4/2986
Cardiac failure chronic (Cardiac disorders) | 1/3006 | 1/2986
Cardiac failure congestive (Cardiac disorders) | 42/3006 | 27/2986
Cardiac tamponade (Cardiac disorders) | 0/3006 | 1/2986
Cardiac valve disease (Cardiac disorders) | 1/3006 | 0/2986
Cardiac ventricular disorder (Cardiac disorders) | 1/3006 | 0/2986
Cardio-respiratory arrest (Cardiac disorders) | 7/3006 | 6/2986
Cardiogenic shock (Cardiac disorders) | 3/3006 | 4/2986
Cardiomegaly (Cardiac disorders) | 1/3006 | 1/2986
Cardiomyopathy (Cardiac disorders) | 3/3006 | 2/2986
Cardiopulmonary failure (Cardiac disorders) | 12/3006 | 10/2986
Conduction disorder (Cardiac disorders) | 0/3006 | 1/2986
Cor pulmonale (Cardiac disorders) | 15/3006 | 12/2986
Cor pulmonale acute (Cardiac disorders) | 2/3006 | 2/2986
Cor pulmonale chronic (Cardiac disorders) | 2/3006 | 4/2986
Coronary artery disease (Cardiac disorders) | 32/3006 | 20/2986
Coronary artery embolism (Cardiac disorders) | 0/3006 | 1/2986
Coronary artery insufficiency (Cardiac disorders) | 1/3006 | 1/2986
Coronary artery occlusion (Cardiac disorders) | 1/3006 | 1/2986
Coronary artery restenosis (Cardiac disorders) | 0/3006 | 1/2986
Coronary artery stenosis (Cardiac disorders) | 6/3006 | 4/2986
Coronary artery thrombosis (Cardiac disorders) | 1/3006 | 0/2986
Diastolic dysfunction (Cardiac disorders) | 0/3006 | 1/2986
Extrasystoles (Cardiac disorders) | 0/3006 | 1/2986
Hypertensive cardiomyopathy (Cardiac disorders) | 0/3006 | 1/2986
Hypertensive heart disease (Cardiac disorders) | 1/3006 | 0/2986
Intracardiac thrombus (Cardiac disorders) | 1/3006 | 0/2986
Ischaemic cardiomyopathy (Cardiac disorders) | 3/3006 | 2/2986
Left ventricular dysfunction (Cardiac disorders) | 2/3006 | 1/2986
Left ventricular failure (Cardiac disorders) | 5/3006 | 6/2986
Mitral valve incompetence (Cardiac disorders) | 3/3006 | 2/2986
Myocardial infarction (Cardiac disorders) | 84/3006 | 65/2986
Myocardial ischaemia (Cardiac disorders) | 13/3006 | 10/2986
Myocarditis (Cardiac disorders) | 1/3006 | 0/2986
Palpitations (Cardiac disorders) | 2/3006 | 2/2986
Pericardial haemorrhage (Cardiac disorders) | 2/3006 | 0/2986
Pericarditis (Cardiac disorders) | 1/3006 | 0/2986
Right ventricular failure (Cardiac disorders) | 6/3006 | 4/2986
Sick sinus syndrome (Cardiac disorders) | 1/3006 | 0/2986
Supraventricular extrasystoles (Cardiac disorders) | 1/3006 | 0/2986
Supraventricular tachycardia (Cardiac disorders) | 8/3006 | 8/2986
Tachyarrhythmia (Cardiac disorders) | 2/3006 | 5/2986
Tachycardia (Cardiac disorders) | 6/3006 | 4/2986
Torsade de pointes (Cardiac disorders) | 1/3006 | 0/2986
Tricuspid valve incompetence (Cardiac disorders) | 0/3006 | 1/2986
Ventricular arrhythmia (Cardiac disorders) | 1/3006 | 1/2986
Ventricular extrasystoles (Cardiac disorders) | 0/3006 | 1/2986
Ventricular fibrillation (Cardiac disorders) | 9/3006 | 3/2986
Ventricular hypokinesia (Cardiac disorders) | 1/3006 | 0/2986
Ventricular tachycardia (Cardiac disorders) | 7/3006 | 7/2986
Adenomatous polyposis coli (Congenital, familial and genetic disorders) | 1/3006 | 0/2986
Arteriovenous malformation (Congenital, familial and genetic disorders) | 0/3006 | 1/2986
Atrial septal defect (Congenital, familial and genetic disorders) | 1/3006 | 0/2986
Congenital myopathy (Congenital, familial and genetic disorders) | 1/3006 | 0/2986
Dermoid cyst (Congenital, familial and genetic disorders) | 0/3006 | 1/2986
Dolichocolon (Congenital, familial and genetic disorders) | 0/3006 | 1/2986
Gastrointestinal angiodysplasia (Congenital, familial and genetic disorders) | 0/3006 | 1/2986
Gastrointestinal angiodysplasia haemorrhagic (Congenital, familial and genetic disorders) | 1/3006 | 0/2986
Gastrointestinal arteriovenous malformation (Congenital, familial and genetic disorders) | 1/3006 | 1/2986
Hydrocele (Congenital, familial and genetic disorders) | 0/3006 | 2/2986
Neurofibromatosis (Congenital, familial and genetic disorders) | 0/3006 | 1/2986
Phimosis (Congenital, familial and genetic disorders) | 1/3006 | 1/2986
Pyloric stenosis (Congenital, familial and genetic disorders) | 0/3006 | 1/2986
Deafness (Ear and labyrinth disorders) | 1/3006 | 0/2986
Hypoacusis (Ear and labyrinth disorders) | 1/3006 | 0/2986
Otosclerosis (Ear and labyrinth disorders) | 1/3006 | 0/2986
Sudden hearing loss (Ear and labyrinth disorders) | 0/3006 | 1/2986
Vertigo (Ear and labyrinth disorders) | 8/3006 | 8/2986
Vertigo positional (Ear and labyrinth disorders) | 0/3006 | 2/2986
Vestibular disorder (Ear and labyrinth disorders) | 1/3006 | 0/2986
Adrenal insufficiency (Endocrine disorders) | 0/3006 | 1/2986
Adrenal mass (Endocrine disorders) | 0/3006 | 1/2986
Diabetes insipidus (Endocrine disorders) | 1/3006 | 0/2986
Hyperparathyroidism (Endocrine disorders) | 2/3006 | 0/2986
Hyperthyroidism (Endocrine disorders) | 2/3006 | 1/2986
Thyroid disorder (Endocrine disorders) | 0/3006 | 1/2986
Amaurosis fugax (Eye disorders) | 1/3006 | 0/2986
Blindness unilateral (Eye disorders) | 0/3006 | 1/2986
Cataract (Eye disorders) | 21/3006 | 23/2986
Conjunctivitis (Eye disorders) | 1/3006 | 0/2986
Eye haemorrhage (Eye disorders) | 0/3006 | 1/2986
Eye pain (Eye disorders) | 0/3006 | 1/2986
Glaucoma (Eye disorders) | 1/3006 | 2/2986
Iridocele (Eye disorders) | 0/3006 | 1/2986
Optic ischaemic neuropathy (Eye disorders) | 1/3006 | 0/2986
Retinal detachment (Eye disorders) | 1/3006 | 2/2986
Retinal tear (Eye disorders) | 1/3006 | 0/2986
Retinal vein occlusion (Eye disorders) | 1/3006 | 0/2986
Vision blurred (Eye disorders) | 0/3006 | 1/2986
Visual disturbance (Eye disorders) | 1/3006 | 0/2986
Vitreous haemorrhage (Eye disorders) | 0/3006 | 1/2986
Abdominal adhesions (Gastrointestinal disorders) | 2/3006 | 2/2986
Abdominal discomfort (Gastrointestinal disorders) | 1/3006 | 0/2986
Abdominal distension (Gastrointestinal disorders) | 1/3006 | 0/2986
Abdominal hernia (Gastrointestinal disorders) | 2/3006 | 5/2986
Abdominal pain (Gastrointestinal disorders) | 18/3006 | 18/2986
Abdominal strangulated hernia (Gastrointestinal disorders) | 1/3006 | 0/2986
Appendicitis perforated (Gastrointestinal disorders) | 0/3006 | 2/2986
Ascites (Gastrointestinal disorders) | 3/3006 | 1/2986
Coeliac disease (Gastrointestinal disorders) | 1/3006 | 0/2986
Colitis (Gastrointestinal disorders) | 3/3006 | 0/2986
Colitis ischaemic (Gastrointestinal disorders) | 1/3006 | 1/2986
Colitis ulcerative (Gastrointestinal disorders) | 0/3006 | 1/2986
Colonic polyp (Gastrointestinal disorders) | 4/3006 | 5/2986
Constipation (Gastrointestinal disorders) | 3/3006 | 3/2986
Crohn's disease (Gastrointestinal disorders) | 0/3006 | 1/2986
Dental caries (Gastrointestinal disorders) | 0/3006 | 2/2986
Diarrhoea (Gastrointestinal disorders) | 12/3006 | 5/2986
Diverticular perforation (Gastrointestinal disorders) | 2/3006 | 1/2986
Diverticulum (Gastrointestinal disorders) | 4/3006 | 5/2986
Diverticulum intestinal (Gastrointestinal disorders) | 0/3006 | 1/2986
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1/3006 | 3/2986
Duodenal perforation (Gastrointestinal disorders) | 1/3006 | 0/2986
Duodenal polyp (Gastrointestinal disorders) | 0/3006 | 1/2986
Duodenal ulcer (Gastrointestinal disorders) | 4/3006 | 3/2986
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1/3006 | 0/2986
Duodenitis (Gastrointestinal disorders) | 1/3006 | 1/2986
Dyspepsia (Gastrointestinal disorders) | 1/3006 | 2/2986
Dysphagia (Gastrointestinal disorders) | 3/3006 | 2/2986
Enterocolitis (Gastrointestinal disorders) | 1/3006 | 0/2986
Erosive duodenitis (Gastrointestinal disorders) | 1/3006 | 0/2986
Faecal incontinence (Gastrointestinal disorders) | 1/3006 | 0/2986
Faecaloma (Gastrointestinal disorders) | 2/3006 | 2/2986
Femoral hernia (Gastrointestinal disorders) | 1/3006 | 0/2986
Femoral hernia, obstructive (Gastrointestinal disorders) | 0/3006 | 1/2986
Flatulence (Gastrointestinal disorders) | 1/3006 | 0/2986
Gastric haemorrhage (Gastrointestinal disorders) | 3/3006 | 2/2986
Gastric polyps (Gastrointestinal disorders) | 1/3006 | 1/2986
Gastric ulcer (Gastrointestinal disorders) | 6/3006 | 3/2986
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0/3006 | 1/2986
Gastric varices haemorrhage (Gastrointestinal disorders) | 1/3006 | 0/2986
Gastric volvulus (Gastrointestinal disorders) | 0/3006 | 1/2986
Gastritis (Gastrointestinal disorders) | 5/3006 | 9/2986
Gastritis erosive (Gastrointestinal disorders) | 1/3006 | 3/2986
Gastritis haemorrhagic (Gastrointestinal disorders) | 2/3006 | 1/2986
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 16/3006 | 11/2986
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2/3006 | 2/2986
Gastrooesophagitis (Gastrointestinal disorders) | 1/3006 | 0/2986
Haematemesis (Gastrointestinal disorders) | 4/3006 | 2/2986
Haematochezia (Gastrointestinal disorders) | 2/3006 | 0/2986
Haemorrhoids (Gastrointestinal disorders) | 5/3006 | 2/2986
Hiatus hernia (Gastrointestinal disorders) | 0/3006 | 5/2986
Ileitis (Gastrointestinal disorders) | 1/3006 | 0/2986
Ileus (Gastrointestinal disorders) | 7/3006 | 9/2986
Ileus paralytic (Gastrointestinal disorders) | 1/3006 | 1/2986
Inguinal hernia (Gastrointestinal disorders) | 21/3006 | 20/2986
Inguinal hernia, obstructive (Gastrointestinal disorders) | 0/3006 | 1/2986
Internal hernia (Gastrointestinal disorders) | 1/3006 | 0/2986
Intestinal angina (Gastrointestinal disorders) | 1/3006 | 0/2986
Intestinal fistula (Gastrointestinal disorders) | 1/3006 | 0/2986
Intestinal haemorrhage (Gastrointestinal disorders) | 0/3006 | 2/2986
Intestinal infarction (Gastrointestinal disorders) | 1/3006 | 0/2986
Intestinal ischaemia (Gastrointestinal disorders) | 2/3006 | 1/2986
Intestinal mucosal hypertrophy (Gastrointestinal disorders) | 1/3006 | 0/2986
Intestinal obstruction (Gastrointestinal disorders) | 2/3006 | 9/2986
Intestinal perforation (Gastrointestinal disorders) | 1/3006 | 1/2986
Intestinal polyp (Gastrointestinal disorders) | 3/3006 | 1/2986
Intra-abdominal haematoma (Gastrointestinal disorders) | 0/3006 | 1/2986
Irritable bowel syndrome (Gastrointestinal disorders) | 1/3006 | 0/2986
Large intestinal haemorrhage (Gastrointestinal disorders) | 0/3006 | 1/2986
Large intestine perforation (Gastrointestinal disorders) | 1/3006 | 4/2986
Loose tooth (Gastrointestinal disorders) | 1/3006 | 0/2986
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 3/3006 | 1/2986
Malabsorption (Gastrointestinal disorders) | 0/3006 | 1/2986
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0/3006 | 1/2986
Mechanical ileus (Gastrointestinal disorders) | 0/3006 | 1/2986
Melaena (Gastrointestinal disorders) | 7/3006 | 4/2986
Mouth cyst (Gastrointestinal disorders) | 0/3006 | 1/2986
Mouth ulceration (Gastrointestinal disorders) | 0/3006 | 1/2986
Nausea (Gastrointestinal disorders) | 0/3006 | 5/2986
Odynophagia (Gastrointestinal disorders) | 0/3006 | 1/2986
Oesophageal stenosis (Gastrointestinal disorders) | 1/3006 | 1/2986
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1/3006 | 0/2986
Oesophagitis (Gastrointestinal disorders) | 2/3006 | 1/2986
Oesophagitis ulcerative (Gastrointestinal disorders) | 0/3006 | 1/2986
Pancreatic duct obstruction (Gastrointestinal disorders) | 1/3006 | 0/2986
Pancreatitis (Gastrointestinal disorders) | 6/3006 | 5/2986
Pancreatitis acute (Gastrointestinal disorders) | 3/3006 | 3/2986
Pancreatitis chronic (Gastrointestinal disorders) | 0/3006 | 1/2986
Parotid lipomatosis (Gastrointestinal disorders) | 0/3006 | 1/2986
Peptic ulcer (Gastrointestinal disorders) | 1/3006 | 0/2986
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 1/3006 | 0/2986
Peritonitis (Gastrointestinal disorders) | 1/3006 | 4/2986
Pneumoperitoneum (Gastrointestinal disorders) | 0/3006 | 1/2986
Polyp colorectal (Gastrointestinal disorders) | 2/3006 | 0/2986
Rectal discharge (Gastrointestinal disorders) | 0/3006 | 1/2986
Rectal haemorrhage (Gastrointestinal disorders) | 1/3006 | 1/2986
Rectal polyp (Gastrointestinal disorders) | 2/3006 | 1/2986
Reflux oesophagitis (Gastrointestinal disorders) | 0/3006 | 3/2986
Salivary gland calculus (Gastrointestinal disorders) | 0/3006 | 1/2986
Salivary gland mass (Gastrointestinal disorders) | 0/3006 | 1/2986
Small intestinal obstruction (Gastrointestinal disorders) | 4/3006 | 4/2986
Small intestinal perforation (Gastrointestinal disorders) | 0/3006 | 1/2986
Stomach discomfort (Gastrointestinal disorders) | 2/3006 | 0/2986
Stomatitis (Gastrointestinal disorders) | 0/3006 | 1/2986
Subileus (Gastrointestinal disorders) | 4/3006 | 1/2986
Umbilical hernia (Gastrointestinal disorders) | 4/3006 | 2/2986
Umbilical hernia, obstructive (Gastrointestinal disorders) | 1/3006 | 0/2986
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 5/3006 | 3/2986
Varices oesophageal (Gastrointestinal disorders) | 1/3006 | 1/2986
Volvulus (Gastrointestinal disorders) | 0/3006 | 1/2986
Vomiting (Gastrointestinal disorders) | 1/3006 | 5/2986
Accidental death (General disorders) | 0/3006 | 1/2986
Adverse drug reaction (General disorders) | 0/3006 | 1/2986
Asthenia (General disorders) | 6/3006 | 7/2986
Cardiac death (General disorders) | 1/3006 | 0/2986
Chest discomfort (General disorders) | 1/3006 | 1/2986
Chest pain (General disorders) | 19/3006 | 23/2986
Cyst rupture (General disorders) | 1/3006 | 0/2986
Death (General disorders) | 24/3006 | 31/2986
Fatigue (General disorders) | 2/3006 | 2/2986
General physical health deterioration (General disorders) | 5/3006 | 3/2986
Impaired healing (General disorders) | 0/3006 | 2/2986
Influenza like illness (General disorders) | 0/3006 | 1/2986
Multi-organ disorder (General disorders) | 0/3006 | 1/2986
Multi-organ failure (General disorders) | 10/3006 | 6/2986
Multimorbidity (General disorders) | 1/3006 | 0/2986
Non-cardiac chest pain (General disorders) | 20/3006 | 18/2986
Oedema (General disorders) | 14/3006 | 8/2986
Pain (General disorders) | 1/3006 | 2/2986
Perforated ulcer (General disorders) | 1/3006 | 0/2986
Polyp (General disorders) | 1/3006 | 0/2986
Pyrexia (General disorders) | 6/3006 | 9/2986
Sudden cardiac death (General disorders) | 2/3006 | 1/2986
Sudden death (General disorders) | 11/3006 | 10/2986
Ulcer (General disorders) | 0/3006 | 1/2986
Acute hepatic failure (Hepatobiliary disorders) | 1/3006 | 0/2986
Bile duct obstruction (Hepatobiliary disorders) | 0/3006 | 1/2986
Bile duct stone (Hepatobiliary disorders) | 2/3006 | 6/2986
Biliary colic (Hepatobiliary disorders) | 0/3006 | 3/2986
Biliary dyskinesia (Hepatobiliary disorders) | 0/3006 | 1/2986
Cholangitis (Hepatobiliary disorders) | 2/3006 | 1/2986
Cholangitis acute (Hepatobiliary disorders) | 0/3006 | 1/2986
Cholecystitis (Hepatobiliary disorders) | 5/3006 | 7/2986
Cholecystitis acute (Hepatobiliary disorders) | 4/3006 | 6/2986
Cholecystitis chronic (Hepatobiliary disorders) | 1/3006 | 1/2986
Cholelithiasis (Hepatobiliary disorders) | 18/3006 | 11/2986
Cholelithiasis obstructive (Hepatobiliary disorders) | 1/3006 | 0/2986
Cholestasis (Hepatobiliary disorders) | 2/3006 | 0/2986
Chronic hepatitis (Hepatobiliary disorders) | 1/3006 | 0/2986
Gallbladder disorder (Hepatobiliary disorders) | 1/3006 | 0/2986
Hepatic cirrhosis (Hepatobiliary disorders) | 0/3006 | 3/2986
Hepatic failure (Hepatobiliary disorders) | 1/3006 | 2/2986
Hepatic function abnormal (Hepatobiliary disorders) | 1/3006 | 0/2986
Hepatitis (Hepatobiliary disorders) | 1/3006 | 0/2986
Hepatitis acute (Hepatobiliary disorders) | 1/3006 | 0/2986
Hepatitis alcoholic (Hepatobiliary disorders) | 2/3006 | 1/2986
Hepatomegaly (Hepatobiliary disorders) | 1/3006 | 0/2986
Jaundice (Hepatobiliary disorders) | 1/3006 | 0/2986
Jaundice cholestatic (Hepatobiliary disorders) | 0/3006 | 1/2986
Anaphylactic reaction (Immune system disorders) | 0/3006 | 1/2986
Anaphylactic shock (Immune system disorders) | 1/3006 | 0/2986
Food allergy (Immune system disorders) | 1/3006 | 1/2986
Hypersensitivity (Immune system disorders) | 0/3006 | 2/2986
Abdominal infection (Infections and infestations) | 1/3006 | 0/2986
Abdominal sepsis (Infections and infestations) | 0/3006 | 1/2986
Abdominal wall abscess (Infections and infestations) | 1/3006 | 0/2986
Abscess (Infections and infestations) | 0/3006 | 1/2986
Abscess intestinal (Infections and infestations) | 1/3006 | 0/2986
Abscess limb (Infections and infestations) | 1/3006 | 1/2986
Appendiceal abscess (Infections and infestations) | 0/3006 | 1/2986
Appendicitis (Infections and infestations) | 2/3006 | 9/2986
Arthritis infective (Infections and infestations) | 1/3006 | 1/2986
Bacteraemia (Infections and infestations) | 1/3006 | 2/2986
Bacterial infection (Infections and infestations) | 0/3006 | 1/2986
Biliary tract infection (Infections and infestations) | 1/3006 | 0/2986
Cellulitis (Infections and infestations) | 12/3006 | 9/2986
Cholecystitis infective (Infections and infestations) | 0/3006 | 1/2986
Clostridial infection (Infections and infestations) | 0/3006 | 1/2986
Clostridium difficile colitis (Infections and infestations) | 3/3006 | 1/2986
Corynebacterium infection (Infections and infestations) | 0/3006 | 1/2986
Cystitis escherichia (Infections and infestations) | 0/3006 | 1/2986
Dengue fever (Infections and infestations) | 0/3006 | 1/2986
Dermo-hypodermitis (Infections and infestations) | 1/3006 | 0/2986
Device related infection (Infections and infestations) | 0/3006 | 1/2986
Diverticulitis (Infections and infestations) | 8/3006 | 7/2986
Empyema (Infections and infestations) | 0/3006 | 2/2986
Endocarditis (Infections and infestations) | 0/3006 | 1/2986
Enterococcal sepsis (Infections and infestations) | 1/3006 | 0/2986
Erysipelas (Infections and infestations) | 0/3006 | 5/2986
Escherichia sepsis (Infections and infestations) | 0/3006 | 1/2986
Fungaemia (Infections and infestations) | 1/3006 | 1/2986
Fungal infection (Infections and infestations) | 0/3006 | 1/2986
Gangrene (Infections and infestations) | 3/3006 | 0/2986
Gastritis viral (Infections and infestations) | 1/3006 | 0/2986
Gastroenteritis (Infections and infestations) | 3/3006 | 5/2986
Gastroenteritis Escherichia coli (Infections and infestations) | 1/3006 | 0/2986
Gastroenteritis salmonella (Infections and infestations) | 0/3006 | 2/2986
Gastroenteritis viral (Infections and infestations) | 1/3006 | 0/2986
Groin abscess (Infections and infestations) | 1/3006 | 1/2986
Haemorrhoid infection (Infections and infestations) | 1/3006 | 0/2986
Helicobacter infection (Infections and infestations) | 0/3006 | 1/2986
Herpes zoster (Infections and infestations) | 1/3006 | 0/2986
Herpes zoster infection neurological (Infections and infestations) | 1/3006 | 0/2986
Hydrocele male infected (Infections and infestations) | 0/3006 | 1/2986
Incision site infection (Infections and infestations) | 1/3006 | 0/2986
Infection (Infections and infestations) | 0/3006 | 1/2986
Intertrigo candida (Infections and infestations) | 1/3006 | 0/2986
Intervertebral discitis (Infections and infestations) | 1/3006 | 0/2986
Joint abscess (Infections and infestations) | 0/3006 | 1/2986
Klebsiella sepsis (Infections and infestations) | 0/3006 | 1/2986
Localised infection (Infections and infestations) | 0/3006 | 1/2986
Meningitis (Infections and infestations) | 0/3006 | 2/2986
Meningitis listeria (Infections and infestations) | 1/3006 | 0/2986
Meningococcal bacteraemia (Infections and infestations) | 0/3006 | 1/2986
Mycobacterial infection (Infections and infestations) | 0/3006 | 1/2986
Necrotising fasciitis (Infections and infestations) | 1/3006 | 1/2986
Neutropenic sepsis (Infections and infestations) | 0/3006 | 1/2986
Nosocomial infection (Infections and infestations) | 1/3006 | 0/2986
Oesophageal candidiasis (Infections and infestations) | 0/3006 | 1/2986
Orchitis (Infections and infestations) | 1/3006 | 1/2986
Oropharyngeal candidiasis (Infections and infestations) | 2/3006 | 0/2986
Osteomyelitis (Infections and infestations) | 1/3006 | 3/2986
Otitis media (Infections and infestations) | 0/3006 | 1/2986
Parotitis (Infections and infestations) | 0/3006 | 1/2986
Perianal abscess (Infections and infestations) | 0/3006 | 1/2986
Periodontal infection (Infections and infestations) | 0/3006 | 1/2986
Periorbital cellulitis (Infections and infestations) | 1/3006 | 0/2986
Perirectal abscess (Infections and infestations) | 1/3006 | 0/2986
Peritoneal abscess (Infections and infestations) | 0/3006 | 1/2986
Peritoneal infection (Infections and infestations) | 1/3006 | 0/2986
Pneumococcal sepsis (Infections and infestations) | 1/3006 | 0/2986
Post procedural infection (Infections and infestations) | 0/3006 | 1/2986
Post procedural pneumonia (Infections and infestations) | 1/3006 | 0/2986
Postoperative wound infection (Infections and infestations) | 2/3006 | 3/2986
Pseudomonas infection (Infections and infestations) | 1/3006 | 0/2986
Sepsis (Infections and infestations) | 26/3006 | 16/2986
Sepsis syndrome (Infections and infestations) | 1/3006 | 2/2986
Septic shock (Infections and infestations) | 11/3006 | 9/2986
Skin infection (Infections and infestations) | 2/3006 | 0/2986
Staphylococcal infection (Infections and infestations) | 1/3006 | 2/2986
Staphylococcal sepsis (Infections and infestations) | 1/3006 | 1/2986
Subcutaneous abscess (Infections and infestations) | 0/3006 | 1/2986
Toxic shock syndrome (Infections and infestations) | 0/3006 | 1/2986
Tuberculosis (Infections and infestations) | 4/3006 | 4/2986
Urinary tract infection (Infections and infestations) | 17/3006 | 24/2986
Urosepsis (Infections and infestations) | 3/3006 | 1/2986
Wound infection (Infections and infestations) | 1/3006 | 2/2986
Wound infection staphylococcal (Infections and infestations) | 0/3006 | 1/2986
Wound sepsis (Infections and infestations) | 1/3006 | 0/2986
Abdominal injury (Injury, poisoning and procedural complications) | 0/3006 | 1/2986
Accident (Injury, poisoning and procedural complications) | 0/3006 | 3/2986
Acetabulum fracture (Injury, poisoning and procedural complications) | 0/3006 | 1/2986
Alcohol poisoning (Injury, poisoning and procedural complications) | 4/3006 | 3/2986
Anaemia postoperative (Injury, poisoning and procedural complications) | 1/3006 | 0/2986
Anastomotic stenosis (Injury, poisoning and procedural complications) | 0/3006 | 1/2986
Ankle fracture (Injury, poisoning and procedural complications) | 5/3006 | 6/2986
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1/3006 | 0/2986
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 1/3006 | 0/2986
Back injury (Injury, poisoning and procedural complications) | 1/3006 | 0/2986
Bladder injury (Injury, poisoning and procedural complications) | 1/3006 | 0/2986
Brain contusion (Injury, poisoning and procedural complications) | 1/3006 | 1/2986
Brain herniation (Injury, poisoning and procedural complications) | 0/3006 | 1/2986
Burn of internal organs (Injury, poisoning and procedural complications) | 0/3006 | 1/2986
Bursa injury (Injury, poisoning and procedural complications) | 1/3006 | 0/2986
Cardiac pacemaker malfunction (Injury, poisoning and procedural complications) | 1/3006 | 0/2986
Caustic injury (Injury, poisoning and procedural complications) | 0/3006 | 1/2986
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0/3006 | 4/2986
Chest injury (Injury, poisoning and procedural complications) | 0/3006 | 1/2986
Concussion (Injury, poisoning and procedural complications) | 2/3006 | 7/2986
Contusion (Injury, poisoning and procedural complications) | 3/3006 | 5/2986
Decerebration (Injury, poisoning and procedural complications) | 0/3006 | 1/2986
Delayed recovery from anaesthesia (Injury, poisoning and procedural complications) | 1/3006 | 0/2986
Device failure (Injury, poisoning and procedural complications) | 0/3006 | 1/2986
Device malfunction (Injury, poisoning and procedural complications) | 0/3006 | 1/2986
Dislocation of joint prosthesis (Injury, poisoning and procedural complications) | 1/3006 | 1/2986
Drug toxicity (Injury, poisoning and procedural complications) | 4/3006 | 1/2986
Face injury (Injury, poisoning and procedural complications) | 1/3006 | 1/2986
Facial bones fracture (Injury, poisoning and procedural complications) | 3/3006 | 2/2986
Fall (Injury, poisoning and procedural complications) | 12/3006 | 19/2986
Femoral neck fracture (Injury, poisoning and procedural complications) | 5/3006 | 9/2986
Femur fracture (Injury, poisoning and procedural complications) | 6/3006 | 7/2986
Fibula fracture (Injury, poisoning and procedural complications) | 2/3006 | 0/2986
Foot fracture (Injury, poisoning and procedural complications) | 1/3006 | 0/2986
Foreign body trauma (Injury, poisoning and procedural complications) | 0/3006 | 2/2986
Fracture (Injury, poisoning and procedural complications) | 1/3006 | 0/2986
Gastrointestinal disorder postoperative (Injury, poisoning and procedural complications) | 0/3006 | 1/2986
Gastrointestinal injury (Injury, poisoning and procedural complications) | 1/3006 | 0/2986
Hand fracture (Injury, poisoning and procedural complications) | 1/3006 | 0/2986
Head injury (Injury, poisoning and procedural complications) | 3/3006 | 1/2986
Hip fracture (Injury, poisoning and procedural complications) | 8/3006 | 9/2986
Humerus fracture (Injury, poisoning and procedural complications) | 3/3006 | 3/2986
Ilium fracture (Injury, poisoning and procedural complications) | 0/3006 | 1/2986
Incision site haemorrhage (Injury, poisoning and procedural complications) | 1/3006 | 0/2986
Incisional hernia (Injury, poisoning and procedural complications) | 2/3006 | 1/2986
Injury (Injury, poisoning and procedural complications) | 0/3006 | 2/2986
Internal injury (Injury, poisoning and procedural complications) | 0/3006 | 1/2986
Joint dislocation (Injury, poisoning and procedural complications) | 1/3006 | 1/2986
Joint injury (Injury, poisoning and procedural complications) | 1/3006 | 1/2986
Joint sprain (Injury, poisoning and procedural complications) | 1/3006 | 0/2986
Limb injury (Injury, poisoning and procedural complications) | 0/3006 | 2/2986
Lower limb fracture (Injury, poisoning and procedural complications) | 0/3006 | 4/2986
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2/3006 | 0/2986
Meniscus lesion (Injury, poisoning and procedural complications) | 2/3006 | 2/2986
Multiple injuries (Injury, poisoning and procedural complications) | 1/3006 | 0/2986
Neck injury (Injury, poisoning and procedural complications) | 1/3006 | 1/2986
Operative haemorrhage (Injury, poisoning and procedural complications) | 0/3006 | 1/2986
Overdose (Injury, poisoning and procedural complications) | 1/3006 | 1/2986
Pacemaker complication (Injury, poisoning and procedural complications) | 0/3006 | 2/2986
Pancreatic injury (Injury, poisoning and procedural complications) | 1/3006 | 0/2986
Patella fracture (Injury, poisoning and procedural complications) | 0/3006 | 1/2986
Pelvic fracture (Injury, poisoning and procedural complications) | 1/3006 | 0/2986
Post gastric surgery syndrome (Injury, poisoning and procedural complications) | 1/3006 | 0/2986
Post procedural bile leak (Injury, poisoning and procedural complications) | 0/3006 | 1/2986
Post procedural fistula (Injury, poisoning and procedural complications) | 0/3006 | 1/2986
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2/3006 | 0/2986
Post-traumatic pain (Injury, poisoning and procedural complications) | 0/3006 | 1/2986
Postoperative ileus (Injury, poisoning and procedural complications) | 3/3006 | 2/2986
Postoperative wound complication (Injury, poisoning and procedural complications) | 1/3006 | 0/2986
Procedural hypotension (Injury, poisoning and procedural complications) | 1/3006 | 1/2986
Pubic rami fracture (Injury, poisoning and procedural complications) | 0/3006 | 1/2986
Radius fracture (Injury, poisoning and procedural complications) | 0/3006 | 2/2986
Rib fracture (Injury, poisoning and procedural complications) | 6/3006 | 9/2986
Road traffic accident (Injury, poisoning and procedural complications) | 1/3006 | 8/2986
Scapula fracture (Injury, poisoning and procedural complications) | 1/3006 | 1/2986
Shunt thrombosis (Injury, poisoning and procedural complications) | 0/3006 | 1/2986
Skin injury (Injury, poisoning and procedural complications) | 0/3006 | 1/2986
Skin laceration (Injury, poisoning and procedural complications) | 3/3006 | 4/2986
Skull fracture (Injury, poisoning and procedural complications) | 1/3006 | 0/2986
Spinal compression fracture (Injury, poisoning and procedural complications) | 6/3006 | 8/2986
Spinal fracture (Injury, poisoning and procedural complications) | 1/3006 | 1/2986
Stent occlusion (Injury, poisoning and procedural complications) | 0/3006 | 1/2986
Stent-graft endoleak (Injury, poisoning and procedural complications) | 1/3006 | 0/2986
Subdural haematoma (Injury, poisoning and procedural complications) | 1/3006 | 1/2986
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0/3006 | 2/2986
Synovial rupture (Injury, poisoning and procedural complications) | 1/3006 | 0/2986
Tendon injury (Injury, poisoning and procedural complications) | 1/3006 | 1/2986
Tendon rupture (Injury, poisoning and procedural complications) | 0/3006 | 3/2986
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 0/3006 | 1/2986
Thermal burn (Injury, poisoning and procedural complications) | 1/3006 | 0/2986
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 2/3006 | 2/2986
Thrombosis in device (Injury, poisoning and procedural complications) | 0/3006 | 1/2986
Tibia fracture (Injury, poisoning and procedural complications) | 2/3006 | 1/2986
Traumatic brain injury (Injury, poisoning and procedural complications) | 0/3006 | 3/2986
Traumatic fracture (Injury, poisoning and procedural complications) | 1/3006 | 0/2986
Ulna fracture (Injury, poisoning and procedural complications) | 0/3006 | 1/2986
Ulnar nerve injury (Injury, poisoning and procedural complications) | 0/3006 | 1/2986
Upper limb fracture (Injury, poisoning and procedural complications) | 1/3006 | 5/2986
Urinary tract injury (Injury, poisoning and procedural complications) | 0/3006 | 1/2986
Vaccination complication (Injury, poisoning and procedural complications) | 1/3006 | 0/2986
Vascular bypass dysfunction (Injury, poisoning and procedural complications) | 1/3006 | 0/2986
Vascular graft occlusion (Injury, poisoning and procedural complications) | 0/3006 | 1/2986
Vena cava injury (Injury, poisoning and procedural complications) | 1/3006 | 0/2986
Wound (Injury, poisoning and procedural complications) | 0/3006 | 1/2986
Wound dehiscence (Injury, poisoning and procedural complications) | 0/3006 | 4/2986
Wound secretion (Injury, poisoning and procedural complications) | 0/3006 | 1/2986
Wrist fracture (Injury, poisoning and procedural complications) | 5/3006 | 2/2986
Blood calcium decreased (Investigations) | 1/3006 | 0/2986
Blood creatine phosphokinase increased (Investigations) | 0/3006 | 1/2986
Blood glucose increased (Investigations) | 1/3006 | 1/2986
Blood pressure increased (Investigations) | 1/3006 | 1/2986
Blood sodium decreased (Investigations) | 0/3006 | 1/2986
Body temperature increased (Investigations) | 0/3006 | 1/2986
C-reactive protein increased (Investigations) | 0/3006 | 1/2986
Cardiac murmur (Investigations) | 0/3006 | 1/2986
Electrocardiogram QT prolonged (Investigations) | 0/3006 | 1/2986
Heart rate irregular (Investigations) | 1/3006 | 1/2986
Hepatic enzyme increased (Investigations) | 0/3006 | 1/2986
International normalised ratio increased (Investigations) | 0/3006 | 1/2986
Investigation (Investigations) | 0/3006 | 5/2986
Oxygen saturation decreased (Investigations) | 1/3006 | 2/2986
Physical examination (Investigations) | 0/3006 | 1/2986
Platelet count decreased (Investigations) | 0/3006 | 1/2986
Prostatic specific antigen increased (Investigations) | 0/3006 | 1/2986
Urine calcium increased (Investigations) | 1/3006 | 0/2986
Urine output decreased (Investigations) | 0/3006 | 1/2986
Weight decreased (Investigations) | 3/3006 | 3/2986
White blood cell count decreased (Investigations) | 0/3006 | 1/2986
White blood cell count increased (Investigations) | 0/3006 | 1/2986
Acidosis (Metabolism and nutrition disorders) | 1/3006 | 0/2986
Anorexia (Metabolism and nutrition disorders) | 0/3006 | 1/2986
Cachexia (Metabolism and nutrition disorders) | 4/3006 | 1/2986
Dehydration (Metabolism and nutrition disorders) | 10/3006 | 14/2986
Diabetes mellitus (Metabolism and nutrition disorders) | 7/3006 | 8/2986
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1/3006 | 3/2986
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 3/3006 | 0/2986
Electrolyte imbalance (Metabolism and nutrition disorders) | 1/3006 | 1/2986
Failure to thrive (Metabolism and nutrition disorders) | 1/3006 | 0/2986
Food intolerance (Metabolism and nutrition disorders) | 0/3006 | 1/2986
Gout (Metabolism and nutrition disorders) | 1/3006 | 2/2986
Hyperglycaemia (Metabolism and nutrition disorders) | 3/3006 | 1/2986
Hyperkalaemia (Metabolism and nutrition disorders) | 3/3006 | 3/2986
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0/3006 | 1/2986
Hypoglycaemia (Metabolism and nutrition disorders) | 4/3006 | 3/2986
Hypokalaemia (Metabolism and nutrition disorders) | 5/3006 | 2/2986
Hypomagnesaemia (Metabolism and nutrition disorders) | 1/3006 | 0/2986
Hyponatraemia (Metabolism and nutrition disorders) | 6/3006 | 5/2986
Hypophosphataemia (Metabolism and nutrition disorders) | 0/3006 | 1/2986
Hypovolaemia (Metabolism and nutrition disorders) | 0/3006 | 1/2986
Malnutrition (Metabolism and nutrition disorders) | 0/3006 | 1/2986
Metabolic acidosis (Metabolism and nutrition disorders) | 1/3006 | 0/2986
Obesity (Metabolism and nutrition disorders) | 0/3006 | 2/2986
Polydipsia (Metabolism and nutrition disorders) | 0/3006 | 1/2986
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0/3006 | 3/2986
Arthralgia (Musculoskeletal and connective tissue disorders) | 2/3006 | 0/2986
Arthritis (Musculoskeletal and connective tissue disorders) | 1/3006 | 3/2986
Back pain (Musculoskeletal and connective tissue disorders) | 10/3006 | 8/2986
Bone cyst (Musculoskeletal and connective tissue disorders) | 0/3006 | 1/2986
Bone pain (Musculoskeletal and connective tissue disorders) | 2/3006 | 1/2986
Bursitis (Musculoskeletal and connective tissue disorders) | 1/3006 | 1/2986
Costochondritis (Musculoskeletal and connective tissue disorders) | 0/3006 | 1/2986
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1/3006 | 2/2986
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 0/3006 | 1/2986
Foot deformity (Musculoskeletal and connective tissue disorders) | 1/3006 | 0/2986
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 0/3006 | 1/2986
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1/3006 | 2/2986
Intervertebral disc displacement (Musculoskeletal and connective tissue disorders) | 0/3006 | 2/2986
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3/3006 | 6/2986
Joint swelling (Musculoskeletal and connective tissue disorders) | 0/3006 | 1/2986
Loose body in joint (Musculoskeletal and connective tissue disorders) | 1/3006 | 0/2986
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1/3006 | 3/2986
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 0/3006 | 1/2986
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2/3006 | 0/2986
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1/3006 | 0/2986
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4/3006 | 7/2986
Myalgia (Musculoskeletal and connective tissue disorders) | 2/3006 | 0/2986
Myalgia intercostal (Musculoskeletal and connective tissue disorders) | 0/3006 | 2/2986
Myopathy steroid (Musculoskeletal and connective tissue disorders) | 0/3006 | 1/2986
Neck pain (Musculoskeletal and connective tissue disorders) | 1/3006 | 0/2986
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 20/3006 | 28/2986
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1/3006 | 3/2986
Osteopenia (Musculoskeletal and connective tissue disorders) | 0/3006 | 1/2986
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1/3006 | 4/2986
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0/3006 | 2/2986
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3/3006 | 1/2986
Pathological fracture (Musculoskeletal and connective tissue disorders) | 3/3006 | 0/2986
Periarthritis (Musculoskeletal and connective tissue disorders) | 0/3006 | 1/2986
Polymyositis (Musculoskeletal and connective tissue disorders) | 0/3006 | 1/2986
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0/3006 | 1/2986
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1/3006 | 1/2986
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 3/3006 | 3/2986
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 2/3006 | 1/2986
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 8/3006 | 3/2986
Spondylitis (Musculoskeletal and connective tissue disorders) | 2/3006 | 0/2986
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1/3006 | 1/2986
Synovial cyst (Musculoskeletal and connective tissue disorders) | 2/3006 | 0/2986
Tendonitis (Musculoskeletal and connective tissue disorders) | 1/3006 | 0/2986
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/3006 | 0/2986
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/3006 | 1/2986
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3/3006 | 3/2986
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/3006 | 0/2986
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/3006 | 0/2986
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/3006 | 1/2986
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 22/3006 | 23/2986
Basosquamous carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/3006 | 0/2986
Basosquamous carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/3006 | 1/2986
Benign colonic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/3006 | 0/2986
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/3006 | 1/2986
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/3006 | 0/2986
Bladder adenocarcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/3006 | 1/2986
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7/3006 | 11/2986
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/3006 | 3/2986
Bladder cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/3006 | 0/2986
Bladder cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/3006 | 0/2986
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6/3006 | 5/2986
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3/3006 | 5/2986
Bone cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/3006 | 0/2986
Bone neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/3006 | 0/2986
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/3006 | 2/2986
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/3006 | 1/2986
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6/3006 | 8/2986
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/3006 | 1/2986
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/3006 | 2/2986
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/3006 | 1/2986
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/3006 | 0/2986
Carcinoid tumour of the small bowel (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/3006 | 0/2986
Carcinoma in situ of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/3006 | 0/2986
Cerebellar tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/3006 | 1/2986
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/3006 | 1/2986
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/3006 | 1/2986
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/3006 | 1/2986
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10/3006 | 11/2986
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/3006 | 1/2986
Colon cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/3006 | 1/2986
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/3006 | 1/2986
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/3006 | 0/2986
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/3006 | 0/2986
Gastric adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/3006 | 1/2986
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7/3006 | 2/2986
Gastric cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/3006 | 0/2986
Gastric cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/3006 | 0/2986
Gastric cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/3006 | 1/2986
Gastric cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/3006 | 1/2986
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3/3006 | 0/2986
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/3006 | 0/2986
Gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/3006 | 1/2986
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/3006 | 0/2986
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/3006 | 0/2986
Head and neck cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/3006 | 2/2986
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/3006 | 2/2986
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3/3006 | 2/2986
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3/3006 | 4/2986
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/3006 | 0/2986
Large intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/3006 | 1/2986
Lentigo maligna stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/3006 | 2/2986
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/3006 | 1/2986
Lip neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/3006 | 1/2986
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/3006 | 0/2986
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/3006 | 0/2986
Lymph node cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/3006 | 1/2986
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/3006 | 0/2986
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/3006 | 0/2986
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/3006 | 2/2986
Malignant melanoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/3006 | 1/2986
Malignant neoplasm of renal pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/3006 | 1/2986
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/3006 | 0/2986
Malignant palate neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/3006 | 1/2986
Malignant pericardial neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/3006 | 1/2986
Malignant respiratory tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/3006 | 1/2986
Malignant urinary tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/3006 | 1/2986
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/3006 | 2/2986
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/3006 | 2/2986
Metastases to adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/3006 | 1/2986
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4/3006 | 7/2986
Metastases to breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/3006 | 1/2986
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4/3006 | 3/2986
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9/3006 | 10/2986
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3/3006 | 4/2986
Metastases to skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/3006 | 1/2986
Metastases to soft tissue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/3006 | 0/2986
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/3006 | 0/2986
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/3006 | 2/2986
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/3006 | 1/2986
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/3006 | 1/2986
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/3006 | 0/2986
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/3006 | 1/2986
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/3006 | 2/2986
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/3006 | 1/2986
Mycosis fungoides (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/3006 | 1/2986
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/3006 | 0/2986
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3/3006 | 1/2986
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3/3006 | 2/2986
Neoplasm recurrence (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/3006 | 2/2986
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/3006 | 1/2986
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/3006 | 4/2986
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/3006 | 2/2986
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/3006 | 4/2986
Oral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/3006 | 1/2986
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/3006 | 1/2986
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3/3006 | 4/2986
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/3006 | 0/2986
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/3006 | 1/2986
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/3006 | 0/2986
Penis carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/3006 | 0/2986
Penis carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/3006 | 1/2986
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 22/3006 | 31/2986
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3/3006 | 0/2986
Prostate cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/3006 | 0/2986
Prostate cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/3006 | 2/2986
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/3006 | 1/2986
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/3006 | 0/2986
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/3006 | 3/2986
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/3006 | 1/2986
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/3006 | 0/2986
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/3006 | 2/2986
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/3006 | 0/2986
Renal cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/3006 | 1/2986
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/3006 | 2/2986
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/3006 | 0/2986
Retroperitoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/3006 | 1/2986
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/3006 | 1/2986
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/3006 | 0/2986
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/3006 | 0/2986
Small cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/3006 | 2/2986
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/3006 | 0/2986
Small intestine carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/3006 | 1/2986
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7/3006 | 5/2986
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/3006 | 5/2986
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/3006 | 1/2986
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/3006 | 0/2986
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/3006 | 1/2986
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3/3006 | 1/2986
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3/3006 | 3/2986
Tumour invasion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/3006 | 0/2986
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/3006 | 1/2986
Altered state of consciousness (Nervous system disorders) | 2/3006 | 2/2986
Amnesia (Nervous system disorders) | 1/3006 | 1/2986
Amyotrophic lateral sclerosis (Nervous system disorders) | 0/3006 | 1/2986
Anoxic encephalopathy (Nervous system disorders) | 1/3006 | 0/2986
Aphasia (Nervous system disorders) | 1/3006 | 0/2986
Brain injury (Nervous system disorders) | 1/3006 | 0/2986
Brain oedema (Nervous system disorders) | 1/3006 | 1/2986
Brain stem infarction (Nervous system disorders) | 0/3006 | 1/2986
Burning sensation (Nervous system disorders) | 0/3006 | 1/2986
Carotid artery disease (Nervous system disorders) | 2/3006 | 1/2986
Carotid artery occlusion (Nervous system disorders) | 3/3006 | 2/2986
Carotid artery stenosis (Nervous system disorders) | 12/3006 | 9/2986
Carpal tunnel syndrome (Nervous system disorders) | 0/3006 | 1/2986
Cerebellar syndrome (Nervous system disorders) | 0/3006 | 1/2986
Cerebral atrophy (Nervous system disorders) | 0/3006 | 1/2986
Cerebral haematoma (Nervous system disorders) | 1/3006 | 0/2986
Cerebral haemorrhage (Nervous system disorders) | 5/3006 | 3/2986
Cerebral infarction (Nervous system disorders) | 7/3006 | 7/2986
Cerebral ischaemia (Nervous system disorders) | 2/3006 | 3/2986
Cerebrovascular accident (Nervous system disorders) | 28/3006 | 28/2986
Cerebrovascular disorder (Nervous system disorders) | 1/3006 | 1/2986
Cervical cord compression (Nervous system disorders) | 0/3006 | 1/2986
Cervical myelopathy (Nervous system disorders) | 0/3006 | 1/2986
Cervicobrachial syndrome (Nervous system disorders) | 0/3006 | 1/2986
Chronic inflammatory demyelinating polyradiculoneuropathy (Nervous system disorders) | 1/3006 | 0/2986
Coma (Nervous system disorders) | 4/3006 | 3/2986
Coma hepatic (Nervous system disorders) | 0/3006 | 1/2986
Complex regional pain syndrome (Nervous system disorders) | 2/3006 | 0/2986
Convulsion (Nervous system disorders) | 5/3006 | 5/2986
Coordination abnormal (Nervous system disorders) | 0/3006 | 1/2986
Dementia (Nervous system disorders) | 1/3006 | 0/2986
Dementia Alzheimer's type (Nervous system disorders) | 0/3006 | 1/2986
Depressed level of consciousness (Nervous system disorders) | 1/3006 | 0/2986
Diabetic coma (Nervous system disorders) | 1/3006 | 0/2986
Dizziness (Nervous system disorders) | 9/3006 | 7/2986
Dysarthria (Nervous system disorders) | 3/3006 | 0/2986
Dyskinesia (Nervous system disorders) | 0/3006 | 1/2986
Embolic stroke (Nervous system disorders) | 0/3006 | 1/2986
Encephalitis (Nervous system disorders) | 1/3006 | 0/2986
Encephalopathy (Nervous system disorders) | 4/3006 | 0/2986
Epilepsy (Nervous system disorders) | 2/3006 | 2/2986
Extrapyramidal disorder (Nervous system disorders) | 0/3006 | 1/2986
Global amnesia (Nervous system disorders) | 1/3006 | 0/2986
Grand mal convulsion (Nervous system disorders) | 2/3006 | 0/2986
Guillain-Barre syndrome (Nervous system disorders) | 1/3006 | 0/2986
Haemorrhage intracranial (Nervous system disorders) | 0/3006 | 1/2986
Haemorrhagic stroke (Nervous system disorders) | 0/3006 | 1/2986
Headache (Nervous system disorders) | 2/3006 | 3/2986
Hemiparesis (Nervous system disorders) | 4/3006 | 2/2986
Hemiplegia (Nervous system disorders) | 1/3006 | 1/2986
Hyperaesthesia (Nervous system disorders) | 1/3006 | 0/2986
Hypercapnic encephalopathy (Nervous system disorders) | 1/3006 | 0/2986
Hypoaesthesia (Nervous system disorders) | 1/3006 | 1/2986
Hypoxic encephalopathy (Nervous system disorders) | 1/3006 | 0/2986
Intercostal neuralgia (Nervous system disorders) | 0/3006 | 1/2986
Intracranial aneurysm (Nervous system disorders) | 0/3006 | 2/2986
Intracranial haematoma (Nervous system disorders) | 1/3006 | 1/2986
Intracranial hypotension (Nervous system disorders) | 1/3006 | 0/2986
Ischaemic cerebral infarction (Nervous system disorders) | 2/3006 | 0/2986
Ischaemic stroke (Nervous system disorders) | 3/3006 | 8/2986
Lethargy (Nervous system disorders) | 1/3006 | 0/2986
Locked-in syndrome (Nervous system disorders) | 0/3006 | 1/2986
Loss of consciousness (Nervous system disorders) | 2/3006 | 0/2986
Mental impairment (Nervous system disorders) | 0/3006 | 2/2986
Migraine (Nervous system disorders) | 1/3006 | 1/2986
Nervous system disorder (Nervous system disorders) | 0/3006 | 1/2986
Neuralgia (Nervous system disorders) | 2/3006 | 0/2986
Neuropathy peripheral (Nervous system disorders) | 3/3006 | 1/2986
Paralysis (Nervous system disorders) | 0/3006 | 1/2986
Paraparesis (Nervous system disorders) | 1/3006 | 1/2986
Paraplegia (Nervous system disorders) | 0/3006 | 1/2986
Paresis (Nervous system disorders) | 2/3006 | 0/2986
Parkinson's disease (Nervous system disorders) | 0/3006 | 1/2986
Polyneuropathy (Nervous system disorders) | 0/3006 | 1/2986
Presyncope (Nervous system disorders) | 2/3006 | 5/2986
Quadriparesis (Nervous system disorders) | 0/3006 | 1/2986
Radicular pain (Nervous system disorders) | 0/3006 | 1/2986
Radiculitis cervical (Nervous system disorders) | 0/3006 | 1/2986
Radiculopathy (Nervous system disorders) | 2/3006 | 0/2986
Ruptured cerebral aneurysm (Nervous system disorders) | 1/3006 | 0/2986
Sciatica (Nervous system disorders) | 0/3006 | 1/2986
Sensory disturbance (Nervous system disorders) | 0/3006 | 1/2986
Somnolence (Nervous system disorders) | 2/3006 | 0/2986
Spinal cord compression (Nervous system disorders) | 2/3006 | 0/2986
Spinal cord infarction (Nervous system disorders) | 0/3006 | 1/2986
Spinal cord ischaemia (Nervous system disorders) | 0/3006 | 1/2986
Status epilepticus (Nervous system disorders) | 2/3006 | 0/2986
Subarachnoid haemorrhage (Nervous system disorders) | 0/3006 | 1/2986
Syncope (Nervous system disorders) | 10/3006 | 13/2986
Syncope vasovagal (Nervous system disorders) | 0/3006 | 1/2986
Transient ischaemic attack (Nervous system disorders) | 12/3006 | 14/2986
Tremor (Nervous system disorders) | 1/3006 | 0/2986
Vertebrobasilar insufficiency (Nervous system disorders) | 3/3006 | 2/2986
Acute psychosis (Psychiatric disorders) | 0/3006 | 1/2986
Agitation (Psychiatric disorders) | 1/3006 | 0/2986
Alcohol abuse (Psychiatric disorders) | 1/3006 | 3/2986
Alcohol withdrawal syndrome (Psychiatric disorders) | 6/3006 | 0/2986
Alcoholism (Psychiatric disorders) | 2/3006 | 0/2986
Anxiety (Psychiatric disorders) | 3/3006 | 1/2986
Completed suicide (Psychiatric disorders) | 2/3006 | 1/2986
Confusional state (Psychiatric disorders) | 1/3006 | 2/2986
Delirium (Psychiatric disorders) | 2/3006 | 1/2986
Depressed mood (Psychiatric disorders) | 1/3006 | 0/2986
Depression (Psychiatric disorders) | 9/3006 | 8/2986
Disorientation (Psychiatric disorders) | 1/3006 | 0/2986
Drug abuse (Psychiatric disorders) | 0/3006 | 1/2986
Drug dependence (Psychiatric disorders) | 2/3006 | 0/2986
Dysthymic disorder (Psychiatric disorders) | 1/3006 | 0/2986
Hallucination, auditory (Psychiatric disorders) | 1/3006 | 0/2986
Insomnia (Psychiatric disorders) | 1/3006 | 0/2986
Major depression (Psychiatric disorders) | 2/3006 | 1/2986
Mental disorder due to a general medical condition (Psychiatric disorders) | 1/3006 | 0/2986
Mental status changes (Psychiatric disorders) | 0/3006 | 2/2986
Neurosis (Psychiatric disorders) | 0/3006 | 1/2986
Nicotine dependence (Psychiatric disorders) | 1/3006 | 1/2986
Panic attack (Psychiatric disorders) | 2/3006 | 1/2986
Psychotic disorder (Psychiatric disorders) | 0/3006 | 1/2986
Suicidal ideation (Psychiatric disorders) | 1/3006 | 1/2986
Suicide attempt (Psychiatric disorders) | 1/3006 | 0/2986
Tobacco withdrawal symptoms (Psychiatric disorders) | 1/3006 | 0/2986
Anuria (Renal and urinary disorders) | 0/3006 | 1/2986
Bladder disorder (Renal and urinary disorders) | 0/3006 | 1/2986
Bladder diverticulum (Renal and urinary disorders) | 1/3006 | 0/2986
Bladder neck obstruction (Renal and urinary disorders) | 1/3006 | 1/2986
Calculus bladder (Renal and urinary disorders) | 1/3006 | 0/2986
Calculus ureteric (Renal and urinary disorders) | 0/3006 | 1/2986
Calculus urinary (Renal and urinary disorders) | 2/3006 | 0/2986
Cystitis noninfective (Renal and urinary disorders) | 1/3006 | 0/2986
Dysuria (Renal and urinary disorders) | 0/3006 | 1/2986
Glomerulonephritis (Renal and urinary disorders) | 1/3006 | 0/2986
Haematuria (Renal and urinary disorders) | 7/3006 | 4/2986
Hydronephrosis (Renal and urinary disorders) | 1/3006 | 5/2986
Nephrolithiasis (Renal and urinary disorders) | 6/3006 | 8/2986
Nephrotic syndrome (Renal and urinary disorders) | 1/3006 | 0/2986
Oliguria (Renal and urinary disorders) | 0/3006 | 1/2986
Renal aneurysm (Renal and urinary disorders) | 1/3006 | 0/2986
Renal artery stenosis (Renal and urinary disorders) | 3/3006 | 1/2986
Renal colic (Renal and urinary disorders) | 0/3006 | 3/2986
Renal cyst (Renal and urinary disorders) | 0/3006 | 1/2986
Renal failure (Renal and urinary disorders) | 7/3006 | 13/2986
Renal failure acute (Renal and urinary disorders) | 16/3006 | 16/2986
Renal failure chronic (Renal and urinary disorders) | 0/3006 | 3/2986
Renal pain (Renal and urinary disorders) | 1/3006 | 1/2986
Renal tubular necrosis (Renal and urinary disorders) | 1/3006 | 0/2986
Stress urinary incontinence (Renal and urinary disorders) | 1/3006 | 0/2986
Urethral disorder (Renal and urinary disorders) | 0/3006 | 1/2986
Urethral obstruction (Renal and urinary disorders) | 0/3006 | 1/2986
Urethral stenosis (Renal and urinary disorders) | 1/3006 | 6/2986
Urinary bladder polyp (Renal and urinary disorders) | 2/3006 | 0/2986
Urinary incontinence (Renal and urinary disorders) | 1/3006 | 1/2986
Urinary retention (Renal and urinary disorders) | 8/3006 | 15/2986
Urinary tract disorder (Renal and urinary disorders) | 0/3006 | 1/2986
Urinary tract obstruction (Renal and urinary disorders) | 1/3006 | 0/2986
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 14/3006 | 20/2986
Calculus prostatic (Reproductive system and breast disorders) | 1/3006 | 0/2986
Cervical dysplasia (Reproductive system and breast disorders) | 0/3006 | 1/2986
Epididymal cyst (Reproductive system and breast disorders) | 0/3006 | 1/2986
Epididymitis (Reproductive system and breast disorders) | 0/3006 | 2/2986
Erectile dysfunction (Reproductive system and breast disorders) | 1/3006 | 1/2986
Menorrhagia (Reproductive system and breast disorders) | 1/3006 | 0/2986
Metrorrhagia (Reproductive system and breast disorders) | 1/3006 | 1/2986
Organic erectile dysfunction (Reproductive system and breast disorders) | 0/3006 | 1/2986
Ovarian cyst (Reproductive system and breast disorders) | 1/3006 | 1/2986
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0/3006 | 1/2986
Prostatic obstruction (Reproductive system and breast disorders) | 1/3006 | 0/2986
Prostatism (Reproductive system and breast disorders) | 2/3006 | 1/2986
Prostatitis (Reproductive system and breast disorders) | 6/3006 | 1/2986
Prostatomegaly (Reproductive system and breast disorders) | 1/3006 | 0/2986
Scrotal oedema (Reproductive system and breast disorders) | 0/3006 | 1/2986
Uterine cyst (Reproductive system and breast disorders) | 1/3006 | 0/2986
Uterine enlargement (Reproductive system and breast disorders) | 0/3006 | 1/2986
Actinomycotic pulmonary infection (Respiratory, thoracic and mediastinal disorders) | 0/3006 | 1/2986
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 6/3006 | 1/2986
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 31/3006 | 29/2986
Alveolitis allergic (Respiratory, thoracic and mediastinal disorders) | 0/3006 | 1/2986
Aspergilloma (Respiratory, thoracic and mediastinal disorders) | 0/3006 | 3/2986
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1/3006 | 1/2986
Asthma (Respiratory, thoracic and mediastinal disorders) | 2/3006 | 0/2986
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2/3006 | 1/2986
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0/3006 | 1/2986
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 3/3006 | 3/2986
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 27/3006 | 35/2986
Bronchopulmonary aspergillosis (Respiratory, thoracic and mediastinal disorders) | 0/3006 | 1/2986
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 3/3006 | 1/2986
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 742/3006 | 688/2986
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5/3006 | 7/2986
Cough (Respiratory, thoracic and mediastinal disorders) | 1/3006 | 2/2986
Cryptogenic organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0/3006 | 1/2986
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 54/3006 | 36/2986
Emphysema (Respiratory, thoracic and mediastinal disorders) | 5/3006 | 9/2986
Foreign body aspiration (Respiratory, thoracic and mediastinal disorders) | 1/3006 | 0/2986
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 10/3006 | 14/2986
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0/3006 | 2/2986
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0/3006 | 1/2986
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1/3006 | 0/2986
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0/3006 | 1/2986
Lower respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 12/3006 | 12/2986
Lung abscess (Respiratory, thoracic and mediastinal disorders) | 2/3006 | 4/2986
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 7/3006 | 1/2986
Lung infection (Respiratory, thoracic and mediastinal disorders) | 3/3006 | 6/2986
Lung infection pseudomonal (Respiratory, thoracic and mediastinal disorders) | 2/3006 | 5/2986
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 2/3006 | 6/2986
Lung injury (Respiratory, thoracic and mediastinal disorders) | 0/3006 | 1/2986
Middle lobe syndrome (Respiratory, thoracic and mediastinal disorders) | 1/3006 | 1/2986
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6/3006 | 4/2986
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 3/3006 | 2/2986
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 3/3006 | 1/2986
Pneumocystis jiroveci pneumonia (Respiratory, thoracic and mediastinal disorders) | 0/3006 | 1/2986
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 4/3006 | 4/2986
Pneumonia klebsiella (Respiratory, thoracic and mediastinal disorders) | 0/3006 | 1/2986
Pneumonia necrotising (Respiratory, thoracic and mediastinal disorders) | 0/3006 | 1/2986
Pneumonia staphylococcal (Respiratory, thoracic and mediastinal disorders) | 3/3006 | 2/2986
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 290/3006 | 296/2986
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2/3006 | 0/2986
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 24/3006 | 26/2986
Pneumothorax traumatic (Respiratory, thoracic and mediastinal disorders) | 1/3006 | 1/2986
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1/3006 | 1/2986
Pseudomonas bronchitis (Respiratory, thoracic and mediastinal disorders) | 0/3006 | 1/2986
Pulmonary bulla (Respiratory, thoracic and mediastinal disorders) | 1/3006 | 0/2986
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0/3006 | 1/2986
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0/3006 | 1/2986
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0/3006 | 1/2986
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 2/3006 | 1/2986
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 5/3006 | 7/2986
Pulmonary tuberculoma (Respiratory, thoracic and mediastinal disorders) | 1/3006 | 0/2986
Pulmonary tuberculosis (Respiratory, thoracic and mediastinal disorders) | 2/3006 | 4/2986
Pyothorax (Respiratory, thoracic and mediastinal disorders) | 1/3006 | 1/2986
Radiation pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1/3006 | 0/2986
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 5/3006 | 3/2986
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 113/3006 | 85/2986
Respiratory fume inhalation disorder (Respiratory, thoracic and mediastinal disorders) | 1/3006 | 1/2986
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1/3006 | 0/2986
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 0/3006 | 1/2986
Tracheobronchitis (Respiratory, thoracic and mediastinal disorders) | 2/3006 | 3/2986
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2/3006 | 0/2986
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0/3006 | 1/2986
Benign lung neoplasm (Respiratory, thoracic and mediastinal disorders) | 0/3006 | 2/2986
Bronchial carcinoma (Respiratory, thoracic and mediastinal disorders) | 9/3006 | 15/2986
Bronchial neoplasm (Respiratory, thoracic and mediastinal disorders) | 2/3006 | 0/2986
Bronchogenic cyst (Respiratory, thoracic and mediastinal disorders) | 0/3006 | 1/2986
Cyanosis (Respiratory, thoracic and mediastinal disorders) | 0/3006 | 1/2986
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 3/3006 | 3/2986
Hypopharyngeal cancer (Respiratory, thoracic and mediastinal disorders) | 1/3006 | 0/2986
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 8/3006 | 12/2986
Large cell carcinoma of the respir. tract stage unspecified (Respiratory, thoracic and mediastinal disorders) | 2/3006 | 3/2986
Laryngeal cancer (Respiratory, thoracic and mediastinal disorders) | 3/3006 | 1/2986
Lung adenocarcinoma (Respiratory, thoracic and mediastinal disorders) | 11/3006 | 6/2986
Lung adenocarcinoma metastatic (Respiratory, thoracic and mediastinal disorders) | 3/3006 | 0/2986
Lung adenocarcinoma recurrent (Respiratory, thoracic and mediastinal disorders) | 0/3006 | 1/2986
Lung cancer metastatic (Respiratory, thoracic and mediastinal disorders) | 4/3006 | 5/2986
Lung carcinoma cell type unspecified recurrent (Respiratory, thoracic and mediastinal disorders) | 0/3006 | 1/2986
Lung carcinoma cell type unspecified stage 0 (Respiratory, thoracic and mediastinal disorders) | 1/3006 | 0/2986
Lung carcinoma cell type unspecified stage III (Respiratory, thoracic and mediastinal disorders) | 1/3006 | 0/2986
Lung neoplasm (Respiratory, thoracic and mediastinal disorders) | 7/3006 | 12/2986
Lung neoplasm malignant (Respiratory, thoracic and mediastinal disorders) | 34/3006 | 40/2986
Lung squamous cell carcinoma stage III (Respiratory, thoracic and mediastinal disorders) | 1/3006 | 0/2986
Lung squamous cell carcinoma stage IV (Respiratory, thoracic and mediastinal disorders) | 1/3006 | 1/2986
Lung squamous cell carcinoma stage unspecified (Respiratory, thoracic and mediastinal disorders) | 6/3006 | 6/2986
Lymphadenopathy mediastinal (Respiratory, thoracic and mediastinal disorders) | 2/3006 | 1/2986
Malignant mediastinal neoplasm (Respiratory, thoracic and mediastinal disorders) | 1/3006 | 1/2986
Malignant pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1/3006 | 1/2986
Mediastinum neoplasm (Respiratory, thoracic and mediastinal disorders) | 0/3006 | 1/2986
Metastases to lung (Respiratory, thoracic and mediastinal disorders) | 2/3006 | 5/2986
Metastatic bronchial carcinoma (Respiratory, thoracic and mediastinal disorders) | 2/3006 | 0/2986
Non-small cell lung cancer (Respiratory, thoracic and mediastinal disorders) | 12/3006 | 10/2986
Non-small cell lung cancer metastatic (Respiratory, thoracic and mediastinal disorders) | 4/3006 | 6/2986
Pharyngeal cancer stage unspecified (Respiratory, thoracic and mediastinal disorders) | 0/3006 | 1/2986
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0/3006 | 1/2986
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 29/3006 | 25/2986
Pulmonary hilum mass (Respiratory, thoracic and mediastinal disorders) | 1/3006 | 0/2986
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2/3006 | 3/2986
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 3/3006 | 1/2986
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0/3006 | 1/2986
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1/3006 | 0/2986
Scoliosis (Respiratory, thoracic and mediastinal disorders) | 1/3006 | 0/2986
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0/3006 | 1/2986
Small cell lung cancer extensive stage (Respiratory, thoracic and mediastinal disorders) | 1/3006 | 1/2986
Small cell lung cancer limited stage (Respiratory, thoracic and mediastinal disorders) | 0/3006 | 1/2986
Small cell lung cancer metastatic (Respiratory, thoracic and mediastinal disorders) | 1/3006 | 4/2986
Small cell lung cancer stage unspecified (Respiratory, thoracic and mediastinal disorders) | 8/3006 | 8/2986
Throat cancer (Respiratory, thoracic and mediastinal disorders) | 1/3006 | 0/2986
Tracheal neoplasm (Respiratory, thoracic and mediastinal disorders) | 1/3006 | 0/2986
Chronic tonsillitis (Respiratory, thoracic and mediastinal disorders) | 1/3006 | 0/2986
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1/3006 | 0/2986
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6/3006 | 4/2986
Influenza (Respiratory, thoracic and mediastinal disorders) | 4/3006 | 5/2986
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0/3006 | 1/2986
Laryngitis (Respiratory, thoracic and mediastinal disorders) | 1/3006 | 1/2986
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0/3006 | 1/2986
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1/3006 | 1/2986
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0/3006 | 2/2986
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1/3006 | 0/2986
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 1/3006 | 0/2986
Oropharyngeal swelling (Respiratory, thoracic and mediastinal disorders) | 0/3006 | 1/2986
Pharyngeal abscess (Respiratory, thoracic and mediastinal disorders) | 1/3006 | 0/2986
Pharyngeal disorder (Respiratory, thoracic and mediastinal disorders) | 1/3006 | 0/2986
Pharyngeal fistula (Respiratory, thoracic and mediastinal disorders) | 0/3006 | 1/2986
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 1/3006 | 1/2986
Pharyngoesophageal diverticulum (Respiratory, thoracic and mediastinal disorders) | 1/3006 | 0/2986
Pharyngolaryngeal abscess (Respiratory, thoracic and mediastinal disorders) | 1/3006 | 0/2986
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0/3006 | 1/2986
Sinus polyp (Respiratory, thoracic and mediastinal disorders) | 0/3006 | 1/2986
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 3/3006 | 7/2986
Tracheal disorder (Respiratory, thoracic and mediastinal disorders) | 0/3006 | 1/2986
Tracheostomy malfunction (Respiratory, thoracic and mediastinal disorders) | 2/3006 | 0/2986
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 13/3006 | 19/2986
Vocal cord paralysis (Respiratory, thoracic and mediastinal disorders) | 0/3006 | 1/2986
Angioedema (Skin and subcutaneous tissue disorders) | 0/3006 | 2/2986
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 4/3006 | 3/2986
Dermal cyst (Skin and subcutaneous tissue disorders) | 1/3006 | 0/2986
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2/3006 | 0/2986
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1/3006 | 0/2986
Eczema (Skin and subcutaneous tissue disorders) | 1/3006 | 2/2986
Parapsoriasis (Skin and subcutaneous tissue disorders) | 1/3006 | 0/2986
Pemphigoid (Skin and subcutaneous tissue disorders) | 1/3006 | 0/2986
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1/3006 | 0/2986
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 1/3006 | 0/2986
Skin ulcer (Skin and subcutaneous tissue disorders) | 2/3006 | 1/2986
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0/3006 | 1/2986
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 2/3006 | 0/2986
Urticaria (Skin and subcutaneous tissue disorders) | 0/3006 | 1/2986
Alcohol use (Social circumstances) | 1/3006 | 0/2986
Social problem (Social circumstances) | 0/3006 | 1/2986
Social stay hospitalisation (Social circumstances) | 2/3006 | 2/2986
Victim of homicide (Social circumstances) | 0/3006 | 1/2986
Adhesiolysis (Surgical and medical procedures) | 0/3006 | 1/2986
Alcohol detoxification (Surgical and medical procedures) | 0/3006 | 1/2986
Appendicectomy (Surgical and medical procedures) | 0/3006 | 1/2986
Arteriovenous fistula operation (Surgical and medical procedures) | 1/3006 | 0/2986
Bladder operation (Surgical and medical procedures) | 1/3006 | 0/2986
Cardiac pacemaker battery replacement (Surgical and medical procedures) | 1/3006 | 0/2986
Cardiac pacemaker insertion (Surgical and medical procedures) | 0/3006 | 1/2986
Cardiac pacemaker replacement (Surgical and medical procedures) | 1/3006 | 1/2986
Cataract operation (Surgical and medical procedures) | 0/3006 | 3/2986
Catheter placement (Surgical and medical procedures) | 1/3006 | 0/2986
Cholecystectomy (Surgical and medical procedures) | 0/3006 | 1/2986
Colectomy (Surgical and medical procedures) | 0/3006 | 1/2986
Coronary angioplasty (Surgical and medical procedures) | 0/3006 | 1/2986
Coronary arterial stent insertion (Surgical and medical procedures) | 0/3006 | 1/2986
Finger amputation (Surgical and medical procedures) | 1/3006 | 1/2986
Gastrointestinal tube insertion (Surgical and medical procedures) | 1/3006 | 0/2986
Hernia repair (Surgical and medical procedures) | 0/3006 | 1/2986
Hip arthroplasty (Surgical and medical procedures) | 1/3006 | 1/2986
Hip surgery (Surgical and medical procedures) | 0/3006 | 1/2986
Hospitalisation (Surgical and medical procedures) | 0/3006 | 1/2986
Ileostomy (Surgical and medical procedures) | 0/3006 | 1/2986
Intervertebral disc operation (Surgical and medical procedures) | 1/3006 | 0/2986
Joint arthroplasty (Surgical and medical procedures) | 0/3006 | 2/2986
Medical device removal (Surgical and medical procedures) | 0/3006 | 1/2986
Nasal polypectomy (Surgical and medical procedures) | 1/3006 | 0/2986
Oxygen supplementation (Surgical and medical procedures) | 1/3006 | 0/2986
Rehabilitation therapy (Surgical and medical procedures) | 1/3006 | 3/2986
Removal of internal fixation (Surgical and medical procedures) | 1/3006 | 0/2986
Respiratory therapy (Surgical and medical procedures) | 0/3006 | 1/2986
Shoulder operation (Surgical and medical procedures) | 0/3006 | 1/2986
Surgery (Surgical and medical procedures) | 1/3006 | 1/2986
Transurethral prostatectomy (Surgical and medical procedures) | 1/3006 | 0/2986
Umbilical hernia repair (Surgical and medical procedures) | 1/3006 | 0/2986
Aortic aneurysm (Vascular disorders) | 11/3006 | 15/2986
Aortic aneurysm rupture (Vascular disorders) | 5/3006 | 3/2986
Aortic disorder (Vascular disorders) | 0/3006 | 1/2986
Aortic dissection (Vascular disorders) | 1/3006 | 0/2986
Aortic occlusion (Vascular disorders) | 0/3006 | 1/2986
Aortic rupture (Vascular disorders) | 1/3006 | 0/2986
Aortic stenosis (Vascular disorders) | 4/3006 | 4/2986
Aortic thrombosis (Vascular disorders) | 0/3006 | 2/2986
Arterial disorder (Vascular disorders) | 1/3006 | 0/2986
Arterial insufficiency (Vascular disorders) | 0/3006 | 1/2986
Arterial occlusive disease (Vascular disorders) | 1/3006 | 4/2986
Arterial thrombosis (Vascular disorders) | 1/3006 | 0/2986
Arterial thrombosis limb (Vascular disorders) | 2/3006 | 1/2986
Arteriosclerosis (Vascular disorders) | 2/3006 | 4/2986
Arteriosclerosis obliterans (Vascular disorders) | 0/3006 | 1/2986
Arteritis (Vascular disorders) | 1/3006 | 1/2986
Bleeding varicose vein (Vascular disorders) | 1/3006 | 0/2986
Cardiovascular insufficiency (Vascular disorders) | 0/3006 | 2/2986
Circulatory collapse (Vascular disorders) | 6/3006 | 1/2986
Deep vein thrombosis (Vascular disorders) | 8/3006 | 14/2986
Embolism (Vascular disorders) | 1/3006 | 0/2986
Femoral artery occlusion (Vascular disorders) | 0/3006 | 4/2986
Haematoma (Vascular disorders) | 5/3006 | 2/2986
Haemorrhage (Vascular disorders) | 0/3006 | 1/2986
Hypertension (Vascular disorders) | 13/3006 | 11/2986
Hypertensive crisis (Vascular disorders) | 2/3006 | 1/2986
Hypotension (Vascular disorders) | 9/3006 | 11/2986
Hypovolaemic shock (Vascular disorders) | 1/3006 | 0/2986
Iliac artery occlusion (Vascular disorders) | 0/3006 | 1/2986
Iliac artery stenosis (Vascular disorders) | 1/3006 | 2/2986
Intermittent claudication (Vascular disorders) | 0/3006 | 6/2986
Ischaemia (Vascular disorders) | 1/3006 | 1/2986
Jugular vein thrombosis (Vascular disorders) | 1/3006 | 0/2986
Orthostatic hypotension (Vascular disorders) | 3/3006 | 5/2986
Peripheral arterial occlusive disease (Vascular disorders) | 2/3006 | 2/2986
Peripheral artery aneurysm (Vascular disorders) | 2/3006 | 1/2986
Peripheral embolism (Vascular disorders) | 1/3006 | 0/2986
Peripheral ischaemia (Vascular disorders) | 0/3006 | 7/2986
Peripheral vascular disorder (Vascular disorders) | 4/3006 | 3/2986
Shock (Vascular disorders) | 4/3006 | 4/2986
Shock haemorrhagic (Vascular disorders) | 2/3006 | 1/2986
Subclavian artery stenosis (Vascular disorders) | 0/3006 | 1/2986
Superior vena caval occlusion (Vascular disorders) | 1/3006 | 1/2986
Thrombophlebitis (Vascular disorders) | 0/3006 | 2/2986
Thrombophlebitis superficial (Vascular disorders) | 0/3006 | 1/2986
Thrombosis (Vascular disorders) | 1/3006 | 6/2986
Varicose ulceration (Vascular disorders) | 1/3006 | 0/2986
Varicose vein (Vascular disorders) | 2/3006 | 0/2986
Vascular shunt (Vascular disorders) | 0/3006 | 1/2986
Venous stasis (Vascular disorders) | 1/3006 | 0/2986
Venous thrombosis (Vascular disorders) | 3/3006 | 1/2986
Venous thrombosis limb (Vascular disorders) | 1/3006 | 2/2986
Wound haemorrhage (Vascular disorders) | 1/3006 | 0/2986
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Placebo | Tiotropium Bromide Inhalation Capsules 18 mcg
Mouth dry (Gastrointestinal disorders) | 80/3006 | 152/2986
Urinary tract infection (Infections and infestations) | 157/3006 | 173/2986
Back pain (Musculoskeletal and connective tissue disorders) | 179/3006 | 190/2986
Headache (Nervous system disorders) | 135/3006 | 169/2986
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 214/3006 | 207/2986
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 1743/3006 | 1706/2986
Cough (Respiratory, thoracic and mediastinal disorders) | 212/3006 | 236/2986
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 404/3006 | 338/2986
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 156/3006 | 157/2986
Influenza (Respiratory, thoracic and mediastinal disorders) | 155/3006 | 153/2986
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 323/3006 | 373/2986
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 157/3006 | 190/2986
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 282/3006 | 285/2986
Hypertension (Vascular disorders) | 273/3006 | 265/2986

LIMITATIONS AND CAVEATS:
Tio patients had significantly longer drug exposure,thus had increased chance of AE.Simple frequencies are biased for AE comparisons;exposure-adjusted incidence rates (IR) should be used. IR for serious AE(>1% patients) are in Outcome Measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.